CLINICAL TRIAL: NCT01638013
Title: Open-label Extension Study in Rheumatoid Arthritis Patients Who Have Completed Phase 2b Study or Phase 3 Study of ASP015K
Brief Title: A Study to Continue ASP015K Treatment to Rheumatoid Arthritis Patients Who Completed Phase IIb Study or Phase III Study of ASP015K
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 015K-CL-RAJ2
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Smyraf; Rheumatoid Arthritis; Peficitinib; ASP015K
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Participants who completed 015K-CL-RAJ1 (Experimental): Participants who completed 015K-CL-RAJ1 (NCT02305849) study and met eligible criteria received starting dose of 50 milligrams (mg) peficitinib tablet orally once daily after breakfast. Dose can be increased to 100mg or 150mg, and decreased to 50mg. For participants who did not have any safety problem, the dose was increased from 50 mg to 100 mg. For participants who did not have any safety problems, and a lack of clinical response (DAS28-ESR >= 3.2 after 4 weeks of peficitinib treatment), dose was increased to 150mg. The treatment was given in this study up to 6 months after peficitinib was approved.
  Interventions: Drug: Peficitinib
- Participants who completed 015K-CL-RAJ3 (Experimental): Participants who completed 015K-CL-RAJ3 (NCT02308163) study and met eligible criteria received 100mg peficitinib tablet orally once daily after breakfast. Dose can be increased to 100mg or 150mg, and decreased to 50mg. For participants who did not have any safety problem, the dose was increased from 50 mg to 100 mg. For participants who did not have any safety problems, and confirmed a lack of clinical response (DAS28-ESR >= 3.2 after 4 weeks of peficitinib treatment), dose was increased to 150mg. The treatment was given in this study up to 6 months after peficitinib was approved.
  Interventions: Drug: Peficitinib
- Participants who completed 015K-CL-RAJ4 (Experimental): Participants who completed 015K-CL-RAJ4 (NCT02305849) study and met eligible criteria received 100mg peficitinib tablet orally once daily after breakfast. Dose can be increased to 100mg or 150mg, and decreased to 50mg. For participants who did not have any safety problem, the dose was increased from 50 mg to 100 mg. For participants who did not have any safety problems, and confirmed a lack of clinical response (DAS28-ESR >= 3.2 after 4 weeks of peficitinib treatment), dose was increased to 150mg. The treatment was given in this study up to 6 months after peficitinib was approved.
  Interventions: Drug: Peficitinib

INTERVENTIONS:
Drug: Peficitinib — Oral Tablet
  Other Names: ASP015K; Smyraf

SUMMARY:
This study evaluated the safety and efficacy of long-term administration of ASP015K in patients who have completed Phase IIb or Phase III studies.

DETAILED DESCRIPTION:
This study was an extension study conducted as an open-label multicenter study in rheumatoid arthritis (RA) participants who completed the Phase IIb Study of ASP015K [015K-CL-RAJ1 (hereinafter referred to as study RAJ1)], Phase III Study of ASP015K [015K-CL-RAJ3 (RAJ3)], or Phase III Study of ASP015K [015K-CL-RAJ4 (RAJ4)]. After the marketing approval in Japan on 26 Mar 2019, this study continued as "post marketing clinical study" in Japan. In Taiwan and Korea, this study continued as "clinical study".

Participants received oral ASP015K once daily (QD) after breakfast. The ASP015K dose was increased later for participants who have no safety problems but showed lack of efficacy.

The duration of treatment with the study drug was differed depending upon the participants.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed treatment with the study drug in studies RAJ1, RAJ3 or RAJ4 as specified in the protocol
* The subject himself/herself wishes to continue taking the study drug, and the investigator or sub-investigator deems continued administration to be necessary or appropriate

Exclusion Criteria:

* There were abnormal findings in the x-ray taken at Week 0, and an acute or chronic infection, tuberculosis infection, or malignancy is suspected
* Hepatitis B virus or hepatitis C virus carrier or has a history of a positive test for human immunodeficiency virus (HIV) infection
* Subject has concurrent autoimmune disease (except Sjogren's syndrome) other than RA or a history of it
* Subject has a clinically significant infection or disease (requiring hospitalization or parenteral therapy)
* Subject has QTc < 300 msec on ECG measurements performed at the study site at Week 52 of studies RAJ3 or RAJ4 and has QTc < 300 msec at retest.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2012-06-13 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (175):
- Japan (159):
  - JP00037, Nagoya, Aichi-ken
  - JP00109, Nagoya, Aichi-ken
  - JP00130, Nagoya, Aichi-ken
  - JP00175, Nagoya, Aichi-ken
  - JP00066, Okazaki, Aichi-ken
  - JP00140, Toyoake, Aichi-ken
  - JP00108, Toyohashi, Aichi-ken
  - JP00170, Toyohashi, Aichi-ken
  - JP00156, Toyota, Aichi-ken
  - JP00068, Yatomi, Aichi-ken
  - JP00180, Asahi, Chiba
  - JP00166, Funabashi, Chiba
  - JP00102, Kamagaya, Chiba
  - JP00115, Narashino, Chiba
  - JP00138, Yotsukaidō, Chiba
  - JP00120, Iizuka, Fukuoka
  - JP00040, Kitakyushu, Fukuoka
  - JP00119, Kitakyushu, Fukuoka
  - JP00071, Kurume, Fukuoka
  - JP00106, Kurume, Fukuoka
  - JP00033, Takasaki, Gunma
  - JP00163, Higashihiroshima, Hiroshima
  - JP00124, Tomakomai, Hokaido
  - JP00026, Asahikawa, Hokkaido
  - JP00090, Hakodate, Hokkaido
  - JP00172, Kitami, Hokkaido
  - JP00125, Kushiro, Hokkaido
  - JP00001, Sapporo, Hokkaido
  - JP00002, Sapporo, Hokkaido
  - JP00003, Sapporo, Hokkaido
  - JP00031, Sapporo, Hokkaido
  - JP00038, Sapporo, Hokkaido
  - JP00114, Sapporo, Hokkaido
  - JP00158, Sapporo, Hokkaido
  - JP00056, Akashi, Hyōgo
  - JP00069, Himeji, Hyōgo
  - JP00136, Itami, Hyōgo
  - JP00041, Katō, Hyōgo
  - JP00012, Kobe, Hyōgo
  - JP00042, Kobe, Hyōgo
  - JP00092, Kobe, Hyōgo
  - JP00154, Kobe, Hyōgo
  - JP00171, Kobe, Hyōgo
  - JP00117, Nishinomiya, Hyōgo
  - JP00107, Hitachi, Ibaraki
  - JP00181, Hitachi-Naka, Ibaraki
  - JP00073, Koga, Ibaraki
  - JP00054, Mito, Ibaraki
  - JP00039, Tsukuba, Ibaraki
  - JP00034, Komatsu, Ishikawa-ken
  - JP00179, Komatsu, Ishikawa-ken
  - JP00028, Morioka, Iwate
  - JP00049, Morioka, Iwate
  - JP00088, Kida-gun, Kagawa-ken
  - JP00084, Isehara, Kanagawa
  - JP00058, Kawasaki, Kanagawa
  - JP00141, Sagamihara, Kanagawa
  - JP00096, Yokohama, Kanagawa
  - JP00045, Zushi, Kanagawa
  - JP00019, Kōshi, Kumamoto
  - JP00057, Tamana, Kumamoto
  - JP00168, Yokkaichi, Mie-ken
  - JP00023, Miyagi-gun, Miyagi
  - JP00169, Ōsaki, Miyagi
  - JP00004, Sendai, Miyagi
  - JP00027, Sendai, Miyagi
  - JP00036, Sendai, Miyagi
  - JP00105, Sendai, Miyagi
  - JP00151, Sendai, Miyagi
  - JP00050, Hyūga, Miyazaki
  - JP00129, Matsumoto, Nagano
  - JP00162, Isehaya, Nagasaki
  - JP00101, Ōmura, Nagasaki
  - JP00103, Ōmura, Nagasaki
  - JP00153, Sasebo, Nagasaki
  - JP00094, Kashihara, Nara
  - JP00025, Nagaoka, Niigata
  - JP00144, Shibata, Niigata
  - JP00064, Beppu, Oita Prefecture
  - JP00051, Setouchi, Okayama-ken
  - JP00011, Hannan, Osaka
  - JP00134, Higashiosaka, Osaka
  - JP00078, Kawachi-Nagano, Osaka
  - JP00137, Sakai, Osaka
  - JP00070, Suita, Osaka
  - JP00086, Suita, Osaka
  - JP00146, Suita, Osaka
  - JP00061, Toyonaka, Osaka
  - JP00075, Ureshino, Saga-ken
  - JP00126, Gyōda, Saitama
  - JP00007, Hiki-gun, Saitama
  - JP00060, Kawagoe, Saitama
  - JP00161, Kawagoe, Saitama
  - JP00062, Kawaguchi, Saitama
  - JP00052, Sayama, Saitama
  - JP00008, Tokorozawa, Saitama
  - JP00133, Kakegawa, Shizuoka
  - JP00077, Kanuma, Tochigi
  - JP00145, Shimotsuke, Tochigi
  - JP00024, Bunkyo-ku, Tokyo
  - JP00043, Bunkyo-ku, Tokyo
  - JP00143, Bunkyo-ku, Tokyo
  - JP00149, Bunkyo-ku, Tokyo
  - JP00152, Bunkyo-ku, Tokyo
  - JP00095, Chiyoda-ku, Tokyo
  - JP00099, Chiyoda-ku, Tokyo
  - JP00142, Chuo-ku, Tokyo
  - JP00063, Hachiōji, Tokyo
  - JP00053, Kiyose, Tokyo
  - JP00072, Meguro-ku, Tokyo
  - JP00083, Meguro-ku, Tokyo
  - JP00148, Ōta-ku, Tokyo
  - JP00100, Setagaya-ku, Tokyo
  - JP00081, Shibuya-ku, Tokyo
  - JP00032, Shinjuku-ku, Tokyo
  - JP00021, Sumida-ku, Tokyo
  - JP00010, Takaoka, Toyama
  - JP00155, Nishimuro-gun, Wakayama
  - JP00104, Shimonoseki, Yamaguchi
  - JP00047, Shūnan, Yamaguchi
  - JP00176, Fukui
  - JP00018, Fukuoka
  - JP00020, Fukuoka
  - JP00035, Fukuoka
  - JP00059, Fukuoka
  - JP00076, Fukuoka
  - JP00131, Fukuoka
  - JP00164, Fukuoka
  - JP00165, Fukushima
  - JP00013, Hiroshima
  - JP00014, Hiroshima
  - JP00015, Hiroshima
  - JP00016, Hiroshima
  - JP00055, Hiroshima
  - JP00065, Kagoshima
  - JP00074, Kagoshima
  - JP00167, Kagoshima
  - JP00093, Kochi
  - JP00022, Kumamoto
  - JP00046, Kumamoto
  - JP00085, Kyoto
  - JP00123, Kyoto
  - JP00159, Kyoto
  - JP00122, Miyazaki
  - JP00080, Nagano
  - JP00174, Nagano
  - JP00098, Nagasaki
  - JP00112, Nagasaki
  - JP00147, Nagasaki
  - JP00006, Niigata
  - JP00118, Okayama
  - JP00150, Osaka
  - JP00157, Osaka
  - JP00017, Ōita
  - JP00044, Shizuoka
  - JP00089, Shizuoka
  - JP00135, Shizuoka
  - JP00009, Toyama
  - JP00139, Toyama
- South Korea (9):
  - KR00504, Daegu
  - KR00505, Gwangju
  - KR00506, Incheon
  - KR00508, Jeonju
  - KR00501, Seoul
  - KR00502, Seoul
  - KR00509, Seoul
  - KR00511, Seoul
  - KR00507, Suwon
- Taiwan (7):
  - TW00709, Kaohsiung City
  - TW00710, Taichung
  - TW00712, Tainan
  - TW00701, Taipei
  - TW00702, Taipei
  - TW00711, Taipei
  - TW00703, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Takeuchi T, Tanaka Y, Tanaka S, Kawakami A, Song YW, Chen YH, Rokuda M, Izutsu H, Ushijima S, Kaneko Y. Safety and Effectiveness of Peficitinib (ASP015K) in Patients with Rheumatoid Arthritis: Final Results (32 Months of Mean Peficitinib Treatment) From a Long-Term, Open-Label Extension Study in Japan, Korea, and Taiwan. Rheumatol Ther. 2021 Mar;8(1):425-442. doi: 10.1007/s40744-021-00280-5. Epub 2021 Mar 3. PMID 33656739
- [Derived] Takeuchi T, Tanaka Y, Tanaka S, Kawakami A, Song YW, Chen YH, Rokuda M, Izutsu H, Ushijima S, Kaneko Y, Nakashima Y, Shiomi T, Yamada E. Safety and effectiveness of peficitinib (ASP015K) in patients with rheumatoid arthritis: interim data (22.7 months mean peficitinib treatment) from a long-term, open-label extension study in Japan, Korea, and Taiwan. Arthritis Res Ther. 2020 Mar 12;22(1):47. doi: 10.1186/s13075-020-2125-2. PMID 32164762
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed 015K-CL-RAJ1 (NCT01649999), 015K-CL-RAJ3 (NCT02308163), 015K-CL-RAJ4 (NCT02305849) and met eligible criteria were enrolled in this study. Participants in the etanercept group in study 015K-CL-RAJ3 (NCT01649999) were not included in this study.
Pre-assignment Details: For participants who were on 50mg at the time of peficitinib approval, dose was increased to 100mg. Participants whose dose increment was not possible were discontinued.
Period: Overall Study
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Started | 201 | 225 | 417
Completed | 70 | 147 | 296
Not Completed | 131 | 78 | 121
Not completed — Adverse Event | 36 | 29 | 48
Not completed — Lack of Efficacy | 39 | 11 | 14
Not completed — Protocol Violation | 10 | 7 | 11
Not completed — Met discontinuation criteria | 4 | 0 | 7
Not completed — Subject Lost to Follow up | 1 | 0 | 1
Not completed — Miscellaneous | 25 | 19 | 23
Not completed — Withdrawal of Consent | 16 | 12 | 16
Not completed — Not met inclusion or exclusion criteria | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) : All participants who received at least 1 dose of the study drug and had measurements for any of the efficacy endpoints.
  Data reported is from baseline of preceding study.
Groups:
- Participants Who Completed 015K-CL-RAJ1: Participants who completed 015K-CL-RAJ1 (NCT02305849) study and met eligible criteria received starting dose of 50mg peficitinib tablet orally once daily after breakfast. Dose can be increased to 100mg or 150mg, and decreased to 50mg. For participants who did not have any safety problem, the dose was increased from 50mg to 100 mg. For participants who did not have any safety problems, and a lack of clinical response (DAS28-ESR >= 3.2 after 4 weeks of peficitinib treatment), dose was increased to 150mg. The treatment was given in this study up to 6 months after peficitinib was approved.
- Total: Total of all reporting groups
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4 | Total
Number analyzed (Participants) | 201 | 224 | 412 | 837
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.7 (11.3) | 55.2 (12.8) | 57.2 (11.5) | 55.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 163 | 293 | 614
  Male | 43 | 61 | 119 | 223
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 201 | 224 | 412 | 837
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: Milligram per deciliter] — Higher CRP indicates greater disease activity. Population: FAS population with available data.
  Milligram per deciliter | 2.214 (2.379) | 2.167 (2.000) | 2.476 (2.077) | 2.331 (2.136)
Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: Millimeter per hour (mm/h)] — Higher ESR indicates greater disease activity. Population: FAS population with available data.
  Millimeter per hour (mm/h)
    number analyzed (Participants) | 201 | 223 | 411 | 835
    (all) | 44.8 (22.2) | 47.0 (25.9) | 50.7 (26.2) | 48.3 (25.3)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: Units on a scale] — Participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item was scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Population: FAS population with available data.
  Units on a scale
    number analyzed (Participants) | 201 | 223 | 412 | 836
    (all) | 0.89 (0.63) | 0.93 (0.67) | 1.00 (0.65) | 0.96 (0.65)
Physician's Global Assessment of Arthritis [Mean (Standard Deviation); unit: Units on a scale] — Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm visual analog scale where 0 = very well and 100 = very poorly. Population: FAS population with available data.
  Units on a scale
    number analyzed (Participants) | 201 | 223 | 412 | 836
    (all) | 55.68 (20.66) | 58.52 (19.55) | 59.47 (19.70) | 58.3 (19.93)
Subject's Global Assessment of Arthritis [Mean (Standard Deviation); unit: Units on a scale] — Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain. Population: FAS population with available data.
  Units on a scale
    number analyzed (Participants) | 201 | 223 | 412 | 836
    (all) | 56.15 (25.10) | 57.40 (25.24) | 54.79 (24.94) | 55.81 (25.06)
Subject's Global Assessment of Arthritis Pain [Mean (Standard Deviation); unit: Units on a scale] — The participant assessed his/her own pain severity on a visual analog scale (VAS) of 0-100 mm on the questionnaire form. Higher SGA of pain (100 mm VAS) scores indicated greater activity pain. Population: FAS population with available data.
  Units on a scale
    number analyzed (Participants) | 201 | 223 | 412 | 836
    (all) | 56.12 (24.71) | 56.79 (25.44) | 54.19 (25.63) | 55.35 (25.36)
Swollen Joint Count (66 Joints) [Mean (Standard Deviation); unit: Swollen joint count] — The participants were examined for the swollen joints and the location was confirmed by the investigator who assessed the 66 joints. Higher SJC indicated greater disease activity. Population: FAS population with available data.
  Swollen joint count
    number analyzed (Participants) | 201 | 223 | 412 | 836
    (all) | 12.0 (6.1) | 12.4 (6.7) | 13.1 (6.9) | 12.7 (6.7)
Tender Joint Count (68 Joints) [Mean (Standard Deviation); unit: Tender joint count] — The participants were examined for the tender joints and the location was confirmed by the investigator who assessed the 68 joints. Higher TJC indicated greater disease activity. Population: FAS population with available data.
  Tender joint count
    number analyzed (Participants) | 201 | 223 | 412 | 836
    (all) | 15.1 (9.3) | 15.0 (9.8) | 14.9 (8.9) | 15 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: AE was defined as any untoward medical occurrence in a participant administered a study drug that did not necessarily have a causal relationship to this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a study drug, whether or not related to the study drug.
Time Frame: Baseline up to end of study (EOS) (up to week 376)
Population: Safety Population: All participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Completed 015K-CL-RAJ1: Participants who completed 015K-CL-RAJ1 (NCT02305849) study and met eligible crietria received starting dose of 50mg peficitinib tablet orally once daily after breakfast. Dose can be increased to 100mg or 150mg, and decreased to 50mg. For participants who did not have any safety problem, the dose was increased from 50 mg to 100 mg. For participants who did not have any safety problems, and a lack of clinical response (DAS28-ESR >= 3.2 after 4 weeks of peficitinib treatment), dose was increased to 150mg. The treatment was given in this study up to 6 months after peficitinib was approved.
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 225 | 417
Participants
  Adverse Events (AE) | 193 | 208 | 395
  Drug related AE (DAE) | 175 | 160 | 321
  Deaths | 0 | 1 | 1
  Serious AE (SAE) | 59 | 56 | 84
  Drug Related serious AE (DSAE) | 22 | 37 | 54
  Grade 3 or higher in severity AE | 75 | 73 | 118
  AE leading to permanent discontinuation of study | 50 | 34 | 56
  DAE leading to permanent discontinuation of drug | 30 | 18 | 44
  SAE leading to permanent discontinuation of drug | 23 | 20 | 32
  DSAE leading to permanent discontinuation of drug | 11 | 12 | 27
  AE leading to dose reduction of study drug | 4 | 8 | 6
  DAE leading to dose reduction of study drug | 4 | 8 | 6
  AE leading to temporary discontinuation of drug | 81 | 86 | 191
  DAE leading to temporary discontinuation of drug | 67 | 76 | 158

2. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) C-Reactive Protein (CRP) Response Through Week 372
Description: ACR20 response: greater than or equal to (≥) 20 percent (%) improvement in tender or swollen joint count; and ≥ 20% improvement in at least 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
  EOT was defined as end of treatment i.e, either early termination (ET) or week 372. EOS was defined as end of study i.e. 28days from EOT.
Time Frame: Baseline of preceding study, weeks 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, 312, 324, 336, 348, 360, 372, EOT, EOS
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Groups:
- Participants Who Completed 015K-CL-RAJ1: Participants who completed 015K-CL-RAJ1 (NCT02305849) study and met eligible criteria received starting dose of 50mg peficitinib tablet orally once daily after breakfast. Dose can be increased to 100mg or 150mg, and decreased to 50mg. For participants who did not have any safety problem, the dose was increased from 50 mg to 100 mg. For participants who did not have any safety problems, and a lack of clinical response (DAS28-ESR >= 3.2 after 4 weeks of peficitinib treatment), dose was increased to 150mg. The treatment was given in this study up to 6 months after peficitinib was approved.
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 29.5 | 82.5 | 86.2
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 37.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 42.2 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 47.2 |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | 55.1 | 81.2 | 85.0
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 59.7 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 63.7 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 63.6 | 85.5 | 89.1
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 65.2 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 62.6 |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | 68.0 | 83.9 | 91.9
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 70.2 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 73.0 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 76.1 | 83.7 | 90.2
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 73.2 | 81.7 | 89.0
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 77.3 | 86.3 | 90.0
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 76.4 | 80.6 | 89.9
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 78.1 | 85.0 | 90.6
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 77.4 | 79.3 | 91.0
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 78.5 | 84.5 | 91.1
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 79.4 | 81.0 | 91.4
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 83.3 | 85.6 | 91.9
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 79.0 | 90.0 | 93.4
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 77.6 | 75.7 | 93.4
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 79.8 | 81.0 | 93.5
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 82.9 | 62.5 | 95.5
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 83.2 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 80.8 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 80.6 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 78.9 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 78.9 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 75.6 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 81.4 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 76.2 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 76.5 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 81.0 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 82.8 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 75.5 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 70.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 87.5 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT | 64.7 | 74.6 | 87.9
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 52.5 | 69.2 | 68.5

3. Secondary Outcome: Percentage of Participants With an ACR50-CRP Response Through Week 372
Description: ACR50 response: ≥50% improvement in tender or swollen joint counts and 50% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional ability via a health assessment questionnaire-Disability Index, and 5) C-reactive protein at each visit.
Time Frame: as for outcome 2
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 8.5 | 62.8 | 67.5
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 9.5 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 14.1 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 23.1 |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | 28.3 | 60.1 | 67.4
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 30.1 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 34.7 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 36.9 | 63.8 | 73.1
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 40.8 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 38.0 |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | 41.3 | 65.9 | 74.5
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 42.9 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 46.6 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 48.5 | 67.3 | 75.7
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 49.0 | 64.4 | 77.5
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 55.3 | 66.1 | 79.1
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 52.1 | 63.9 | 75.1
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 54.7 | 64.2 | 77.5
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 56.4 | 64.6 | 77.9
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 56.2 | 67.6 | 76.1
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 59.5 | 72.4 | 78.3
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 63.3 | 68.0 | 77.2
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 62.2 | 75.7 | 74.5
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 64.7 | 70.3 | 78.9
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 61.4 | 71.4 | 76.1
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 63.1 | 62.5 | 77.3
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 68.2 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 61.5 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 64.3 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 61.1 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 62.2 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 63.3 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 65.1 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 61.9 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 63.0 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 59.5 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 62.5 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 60.4 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 50.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 68.8 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT | 45.8 | 59.8 | 73.8
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 31.7 | 41.5 | 47.2

4. Secondary Outcome: Percentage of Participants With an ACR70-CRP Response Through Week 372
Description: ACR70 response: ≥ 70% improvement in tender or swollen joint counts and 70% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional ability via a health assessment questionnaire-Disability Index, and 5) C-reactive protein at each visit.
Time Frame: as for outcome 2
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 3.5 | 42.2 | 45.9
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 4.5 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 6.0 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 9.0 |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | 12.1 | 40.4 | 46.1
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 12.2 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 13.2 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 17.1 | 40.6 | 51.5
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 18.5 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 17.9 |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | 22.7 | 42.4 | 50.9
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 22.6 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 23.9 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 25.2 | 41.3 | 54.8
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 24.2 | 45.5 | 53.7
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 26.7 | 42.6 | 56.7
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 29.3 | 44.4 | 55.3
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 29.9 | 43.9 | 56.0
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 35.3 | 47.6 | 57.3
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 35.4 | 48.6 | 52.6
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 36.5 | 48.3 | 55.4
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 36.7 | 48.5 | 52.9
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 39.5 | 48.6 | 48.1
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 39.7 | 48.6 | 52.6
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 42.1 | 47.6 | 58.7
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 44.1 | 50.0 | 59.1
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 46.7 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 41.3 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 43.9 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 44.2 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 46.7 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 43.3 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 44.2 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 41.7 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 40.7 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 46.8 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 50.0 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 41.5 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 27.5 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 50.0 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0.0 |  |
  EOT | 29.9 | 39.7 | 53.4
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 19.8 | 24.6 | 33.7

5. Secondary Outcome: Percentage of Participants With an ACR20 Erythrocyte Sedimentation Rate (ESR) Response Through Week 372
Description: ACR20 response: ≥20% improvement in tender or swollen joint count; and ≥ 20% improvement in at least 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) ESR at each visit.
Time Frame: as for outcome 2
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 28.5 | 80.3 | 85.7
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 37.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 42.2 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 45.7 |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | 52.0 | 80.7 | 85.3
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 61.2 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 63.2 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 63.6 | 84.5 | 88.8
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 65.2 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 63.1 |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | 66.3 | 82.4 | 91.1
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 67.9 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 70.6 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 74.2 | 82.7 | 88.8
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 73.2 | 81.7 | 88.5
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 76.7 | 84.2 | 90.3
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 74.3 | 80.0 | 89.6
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 77.4 | 83.2 | 90.2
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 75.2 | 79.3 | 90.6
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 76.9 | 83.1 | 90.6
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 77.8 | 80.2 | 90.9
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 81.7 | 84.5 | 91.9
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 77.3 | 90.0 | 91.5
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 77.6 | 73.0 | 90.8
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 80.7 | 81.0 | 93.5
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 80.2 | 62.5 | 95.5
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 82.2 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 78.8 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 80.6 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 76.8 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 77.8 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 74.4 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 79.1 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 73.8 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 75.3 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 78.5 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 79.7 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 75.5 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 65.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 81.3 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT | 64.2 | 74.6 | 87.4
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 53.5 | 67.7 | 68.5

6. Secondary Outcome: Percentage of Participants With an ACR50-ESR Response Through Week 372
Description: ACR50 response: ≥50% improvement in tender or swollen joint counts and 50% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional ability via a health assessment questionnaire-Disability Index, and 5) ESR at each visit.
Time Frame: as for outcome 2
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of Participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of Participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 8.0 | 58.3 | 65.3
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 9.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 13.1 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 21.6 |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | 24.2 | 58.3 | 66.4
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 29.1 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 31.1 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 33.2 | 60.9 | 71.1
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 38.6 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 34.6 |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | 38.4 | 64.4 | 72.2
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 41.1 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 44.8 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 45.4 | 62.2 | 74.1
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 45.9 | 62.8 | 74.7
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 51.3 | 65.0 | 76.8
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 49.3 | 61.7 | 73.7
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 54.7 | 61.8 | 74.6
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 54.9 | 63.4 | 75.3
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 55.4 | 64.9 | 75.6
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 58.7 | 71.6 | 75.4
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 60.8 | 66.0 | 77.2
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 61.3 | 70.0 | 72.6
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 63.8 | 67.6 | 76.3
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 57.9 | 61.9 | 73.9
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 60.4 | 62.5 | 72.7
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 63.6 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 58.7 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 63.3 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 56.8 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 57.8 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 55.6 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 59.3 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 58.3 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 60.5 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 55.7 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 54.7 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 56.6 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 45.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 62.5 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT | 45.8 | 58.9 | 72.3
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 28.7 | 38.5 | 46.1

7. Secondary Outcome: Percentage of Participants With an ACR70-ESR Response Through Week 372
Description: ACR70 response: ≥ 70% improvement in tender or swollen joint counts and 70% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional ability via a health assessment questionnaire-Disability Index, and 5) ESR at each visit.
Time Frame: as for outcome 2
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 2.5 | 36.8 | 41.3
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 4.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 5.5 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 7.0 |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | 10.1 | 36.2 | 42.9
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 9.7 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 11.1 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 12.8 | 36.2 | 47.0
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 16.3 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 17.3 |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | 22.1 | 38.0 | 44.6
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 20.2 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 19.6 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 22.1 | 38.3 | 50.1
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 21.0 | 41.4 | 50.8
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 25.3 | 38.8 | 51.9
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 27.1 | 40.0 | 51.5
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 28.5 | 39.9 | 52.8
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 34.6 | 42.7 | 52.1
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 32.3 | 43.9 | 49.3
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 34.1 | 39.7 | 53.1
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 34.2 | 42.3 | 49.3
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 37.8 | 47.1 | 46.2
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 37.1 | 45.9 | 50.0
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 36.8 | 47.6 | 56.5
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 42.3 | 50.0 | 59.1
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 44.9 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 42.3 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 43.9 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 41.1 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 42.2 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 40.0 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 38.4 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 39.3 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 35.8 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 43.0 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 43.8 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 35.8 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 27.5 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 37.5 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0.0 |  |
  EOT | 28.4 | 38.4 | 50.7
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 17.8 | 20.0 | 32.6

8. Secondary Outcome: Change From Baseline of Preceding Study in DAS28-CRP Through Week 372
Description: DAS28-CRP response consisted of following parameters: TJC (28 joints), SJC (28 joints), CRP, SGA, and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 × SGA + 0.96. DAS28-CRP scores range from 0.96 to approximately 10. Higher DAS28 score indicated greater disease activity.
Time Frame: Baseline of preceding study and weeks 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, 312, 324, 336, 348, 360, 372, EOT, EOS
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 411
  Week 0 | -0.71 (1.10) | -2.67 (1.32) | -2.79 (1.23)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -1.04 (1.10) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -1.09 (1.15) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -1.41 (1.13) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | -1.61 (1.17) | -2.64 (1.34) | -2.82 (1.26)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -1.76 (1.16) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -1.85 (1.19) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | -1.92 (1.18) | -2.66 (1.34) | -2.93 (1.20)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -2.03 (1.16) |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | -1.97 (1.21) |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | -2.08 (1.10) | -2.79 (1.34) | -3.01 (1.16)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -2.12 (1.15) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -2.24 (1.16) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | -2.22 (1.19) | -2.77 (1.31) | -3.08 (1.17)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -2.25 (1.19) | -2.71 (1.37) | -3.06 (1.16)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -2.35 (1.32) | -2.88 (1.34) | -3.13 (1.16)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -2.41 (1.28) | -2.77 (1.37) | -3.12 (1.18)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -2.49 (1.24) | -2.82 (1.35) | -3.16 (1.11)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -2.57 (1.28) | -2.88 (1.41) | -3.22 (1.13)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -2.51 (1.33) | -3.02 (1.33) | -3.17 (1.18)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -2.58 (1.39) | -2.98 (1.48) | -3.19 (1.14)
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | -2.67 (1.25) | -2.96 (1.49) | -3.12 (1.28)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -2.59 (1.28) | -3.15 (1.40) | -3.25 (1.25)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -2.61 (1.27) | -3.06 (1.58) | -3.16 (1.25)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -2.57 (1.37) | -3.14 (1.52) | -3.34 (1.21)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -2.70 (1.32) | -3.14 (1.51) | -3.14 (1.27)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -2.76 (1.17) | -3.52 (NA) — Standard Deviation (SD) not estimable as there is only one participant. | -4.01 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -2.70 (1.38) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -2.75 (1.35) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -2.77 (1.36) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -2.75 (1.42) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -2.75 (1.41) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -2.86 (1.29) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -2.81 (1.39) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -2.81 (1.42) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -2.79 (1.36) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -2.89 (1.29) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -2.65 (1.23) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -2.53 (1.25) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -3.28 (1.06) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -4.63 (NA) — SD not estimable as there is only one participant. |  |
  EOS: number analyzed (Participants) | 201 | 221 | 412
  EOS | -2.14 (1.57) | -2.67 (1.50) | -3.05 (1.30)
  EOT: number analyzed (Participants) | 101 | 65 | 89
  EOT | -1.59 (1.38) | -2.01 (1.41) | -2.13 (1.45)

9. Secondary Outcome: Change From Baseline of Preceding Studies in DAS28-ESR Through Week 372
Description: DAS28-ESR response consisted of following parameters: TJC (28 joints), SJC (28 joints), ESR, SGA, and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 × SGA. DAS28-ESR scores range from 0 to approximately 10. Higher DAS28 score indicated greater disease activity.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
units on a scale
  Week 0: number analyzed (Participants) | 199 | 221 | 410
  Week 0 | -0.70 (1.09) | -2.70 (1.40) | -2.83 (1.30)
  Week 2: number analyzed (Participants) | 199 | 0 | 0
  Week 2 | -1.03 (1.12) |  |
  Week 4: number analyzed (Participants) | 198 | 0 | 0
  Week 4 | -1.11 (1.21) |  |
  Week 8: number analyzed (Participants) | 197 | 0 | 0
  Week 8 | -1.43 (1.12) |  |
  Week 12: number analyzed (Participants) | 197 | 217 | 407
  Week 12 | -1.66 (1.19) | -2.68 (1.41) | -2.90 (1.33)
  Week 16: number analyzed (Participants) | 195 | 0 | 0
  Week 16 | -1.83 (1.21) |  |
  Week 20: number analyzed (Participants) | 189 | 0 | 0
  Week 20 | -1.88 (1.19) |  |
  Week 24: number analyzed (Participants) | 186 | 205 | 392
  Week 24 | -1.96 (1.17) | -2.71 (1.40) | -2.99 (1.29)
  Week 28: number analyzed (Participants) | 182 | 0 | 0
  Week 28 | -2.05 (1.15) |  |
  Week 32: number analyzed (Participants) | 178 | 0 | 0
  Week 32 | -2.03 (1.24) |  |
  Week 36: number analyzed (Participants) | 171 | 204 | 379
  Week 36 | -2.14 (1.16) | -2.85 (1.44) | -3.07 (1.24)
  Week 40: number analyzed (Participants) | 167 | 0 | 0
  Week 40 | -2.18 (1.19) |  |
  Week 44: number analyzed (Participants) | 162 | 0 | 0
  Week 44 | -2.28 (1.18) |  |
  Week 48: number analyzed (Participants) | 162 | 195 | 366
  Week 48 | -2.28 (1.22) | -2.82 (1.42) | -3.13 (1.27)
  Week 60: number analyzed (Participants) | 156 | 190 | 354
  Week 60 | -2.32 (1.26) | -2.78 (1.46) | -3.11 (1.24)
  Week 72: number analyzed (Participants) | 149 | 181 | 348
  Week 72 | -2.39 (1.37) | -2.91 (1.44) | -3.22 (1.28)
  Week 84: number analyzed (Participants) | 138 | 177 | 337
  Week 84 | -2.45 (1.33) | -2.81 (1.46) | -3.20 (1.28)
  Week 96: number analyzed (Participants) | 135 | 171 | 305
  Week 96 | -2.59 (1.32) | -2.84 (1.45) | -3.21 (1.18)
  Week 108: number analyzed (Participants) | 132 | 163 | 266
  Week 108 | -2.64 (1.35) | -2.92 (1.52) | -3.31 (1.25)
  Week 120: number analyzed (Participants) | 129 | 147 | 212
  Week 120 | -2.54 (1.39) | -3.05 (1.48) | -3.26 (1.24)
  Week 132: number analyzed (Participants) | 125 | 114 | 175
  Week 132 | -2.67 (1.44) | -2.98 (1.58) | -3.33 (1.24)
  Week 144: number analyzed (Participants) | 119 | 96 | 135
  Week 144 | -2.76 (1.30) | -3.00 (1.59) | -3.30 (1.36)
  Week 156: number analyzed (Participants) | 118 | 70 | 105
  Week 156 | -2.67 (1.34) | -3.14 (1.52) | -3.32 (1.40)
  Week 168: number analyzed (Participants) | 115 | 37 | 76
  Week 168 | -2.68 (1.32) | -3.13 (1.69) | -3.18 (1.27)
  Week 180: number analyzed (Participants) | 112 | 21 | 45
  Week 180 | -2.64 (1.40) | -3.08 (1.80) | -3.38 (1.31)
  Week 192: number analyzed (Participants) | 109 | 8 | 22
  Week 192 | -2.73 (1.35) | -3.25 (1.52) | -3.11 (1.32)
  Week 204: number analyzed (Participants) | 106 | 1 | 1
  Week 204 | -2.79 (1.20) | -3.04 (NA) — SD not estimable as there is only one participant. | -4.29 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 102 | 0 | 0
  Week 216 | -2.73 (1.32) |  |
  Week 228: number analyzed (Participants) | 97 | 0 | 0
  Week 228 | -2.80 (1.35) |  |
  Week 240: number analyzed (Participants) | 94 | 0 | 0
  Week 240 | -2.83 (1.37) |  |
  Week 252: number analyzed (Participants) | 89 | 0 | 0
  Week 252 | -2.83 (1.38) |  |
  Week 264: number analyzed (Participants) | 89 | 0 | 0
  Week 264 | -2.75 (1.39) |  |
  Week 276: number analyzed (Participants) | 85 | 0 | 0
  Week 276 | -2.84 (1.27) |  |
  Week 288: number analyzed (Participants) | 83 | 0 | 0
  Week 288 | -2.77 (1.35) |  |
  Week 300: number analyzed (Participants) | 80 | 0 | 0
  Week 300 | -2.76 (1.34) |  |
  Week 312: number analyzed (Participants) | 78 | 0 | 0
  Week 312 | -2.77 (1.32) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -2.84 (1.25) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -2.62 (1.29) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -2.52 (1.33) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -3.07 (1.17) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -5.13 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 200 | 222 | 411
  EOT | -2.14 (1.61) | -2.69 (1.62) | -3.11 (1.37)
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | -1.58 (1.43) | -2.00 (1.37) | -2.13 (1.41)

10. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP Score < 2.6 Through Week 372
Description: DAS28-CRP response consisted of following parameters: TJC (28 joints), SJC (28 joints), CRP, SGA, and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 × SGA + 0.96. DAS28-CRP scores range from 0.96 to approximately 10. Higher DAS28 score indicated greater disease activity. DAS28-CRP <2.6 = remission, DAS28-CRP <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity.
Time Frame: Weeks 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, 312, 324, 336, 348, 360, 372, EOT, EOS
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 224 | 411
  Week 0 | 8.0 | 55.4 | 58.2
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 13.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 16.1 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 15.1 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 20.2 | 53.9 | 60.3
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 23.0 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 27.4 |  |
  Week 24: number analyzed (Participants) | 187 | 208 | 394
  Week 24 | 26.2 | 56.3 | 62.2
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 29.9 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 29.1 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 381
  Week 36 | 30.8 | 58.3 | 65.4
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 36.9 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 39.9 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 39.3 | 56.3 | 69.2
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 43.9 | 57.1 | 66.6
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 46.7 | 63.9 | 71.1
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 51.4 | 60.6 | 70.7
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 54.7 | 63.6 | 71.3
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 51.1 | 62.8 | 72.7
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 57.7 | 66.9 | 76.1
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 55.6 | 65.5 | 74.3
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 60.0 | 66.0 | 74.8
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 59.7 | 71.4 | 72.6
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 61.2 | 62.2 | 72.4
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 58.8 | 66.7 | 82.6
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 64.0 | 87.5 | 68.2
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 65.4 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 63.5 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 61.2 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 65.3 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 66.7 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 62.2 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 70.9 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 63.1 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 67.9 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 65.8 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 71.9 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 60.4 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 65.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 81.3 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0.0 |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | 45.3 | 57.2 | 69.4
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 22.8 | 35.4 | 44.9

11. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR Score < 2.6 Through Week 372
Description: DAS28-ESR response consisted of following parameters: TJC (28 joints), SJC (28 joints), ESR, SGA , and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 × SGA. DAS28-ESR scores range from 0 to approximately 10. Higher DAS28 score indicated greater disease activity. DAS28-ESR <2.6 = remission, DAS28-ESR <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity.
Time Frame: as for outcome 10
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 411
  Week 0 | 4.5 | 30.9 | 38.0
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 4.5 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 7.0 |  |
  Week 8: number analyzed (Participants) | 197 | 0 | 0
  Week 8 | 7.6 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 12.1 | 36.1 | 39.7
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 13.3 |  |
  Week 20: number analyzed (Participants) | 189 | 0 | 0
  Week 20 | 12.7 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 393
  Week 24 | 13.9 | 35.3 | 43.3
  Week 28: number analyzed (Participants) | 183 | 0 | 0
  Week 28 | 18.0 |  |
  Week 32: number analyzed (Participants) | 178 | 0 | 0
  Week 32 | 16.9 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 380
  Week 36 | 18.6 | 37.4 | 45.8
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 17.3 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 20.9 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 20.9 | 39.1 | 48.0
  Week 60: number analyzed (Participants) | 157 | 191 | 355
  Week 60 | 22.9 | 36.1 | 45.4
  Week 72: number analyzed (Participants) | 150 | 182 | 349
  Week 72 | 28.7 | 47.3 | 51.6
  Week 84: number analyzed (Participants) | 139 | 178 | 338
  Week 84 | 26.6 | 41.0 | 50.0
  Week 96: number analyzed (Participants) | 136 | 172 | 306
  Week 96 | 34.6 | 39.5 | 48.7
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 32.3 | 47.6 | 52.1
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 31.5 | 46.6 | 49.8
  Week 132: number analyzed (Participants) | 126 | 115 | 175
  Week 132 | 34.9 | 47.8 | 54.3
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 35.0 | 48.5 | 55.6
  Week 156: number analyzed (Participants) | 119 | 70 | 105
  Week 156 | 32.8 | 48.6 | 53.3
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 36.2 | 54.1 | 47.4
  Week 180: number analyzed (Participants) | 113 | 21 | 45
  Week 180 | 33.6 | 38.1 | 55.6
  Week 192: number analyzed (Participants) | 110 | 8 | 22
  Week 192 | 39.1 | 37.5 | 45.5
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 35.5 | 0.0 | 100.0
  Week 216: number analyzed (Participants) | 103 | 0 | 0
  Week 216 | 35.9 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 43.9 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 37.9 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 40.0 |  |
  Week 264: number analyzed (Participants) | 89 | 0 | 0
  Week 264 | 32.6 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 38.4 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 41.7 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 35.8 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 38.0 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 39.1 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 32.1 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 27.5 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 31.3 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0.0 |  |
  EOT | 27.4 | 42.9 | 49.8
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 14.9 | 20.0 | 20.2

12. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP Score <= 3.2 Through Week 372
Description: DAS28-CRP response consisted of following parameters: TJC (28 joints), SJC (28 joints), CRP, SGA, and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 × SGA + 0.96. DAS28-CRP scores range from 0.96 to approximately 10. Higher DAS28 score indicated greater disease activity. DAS28-CRP <2.6 = remission.
Time Frame: as for outcome 10
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 224 | 411
  Week 0 | 18.5 | 73.7 | 72.7
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 24.5 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 25.1 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 33.2 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 38.9 | 73.1 | 74.0
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 42.3 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 46.8 |  |
  Week 24: number analyzed (Participants) | 187 | 208 | 394
  Week 24 | 49.7 | 72.1 | 78.4
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 51.6 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 50.8 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 381
  Week 36 | 56.4 | 75.2 | 79.3
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 59.5 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 60.1 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 61.3 | 75.6 | 82.0
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 64.3 | 75.9 | 83.1
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 64.7 | 79.8 | 84.5
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 68.6 | 79.4 | 83.7
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 75.2 | 80.3 | 86.0
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 77.4 | 78.0 | 87.6
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 74.6 | 85.1 | 86.9
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 77.0 | 84.5 | 87.4
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 81.7 | 82.5 | 86.7
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 78.2 | 80.0 | 85.8
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 76.7 | 78.4 | 86.8
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 75.4 | 81.0 | 89.1
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 76.6 | 87.5 | 90.9
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 83.2 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 75.0 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 82.7 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 80.0 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 77.8 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 82.2 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 86.0 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 83.3 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 82.7 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 83.5 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 84.4 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 77.4 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 80.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 100.0 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | 61.7 | 71.6 | 84.0
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 40.6 | 47.7 | 60.7

13. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR Score <= 3.2 Through Week 372
Description: DAS28-ESR response consisted of following parameters: TJC (28 joints), SJC (28 joints), ESR, SGA, and calculated according to description: DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 × SGA. DAS28-ESR scores range from 0 to approximately 10. Higher DAS28 score indicated greater disease activity. DAS28-ESR <2.6 = remission.
Time Frame: as for outcome 10
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 411
  Week 0 | 8.5 | 56.5 | 55.7
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 13.5 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 14.6 |  |
  Week 8: number analyzed (Participants) | 197 | 0 | 0
  Week 8 | 14.2 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 22.7 | 53.0 | 59.6
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 22.4 |  |
  Week 20: number analyzed (Participants) | 189 | 0 | 0
  Week 20 | 23.8 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 393
  Week 24 | 28.3 | 54.1 | 62.3
  Week 28: number analyzed (Participants) | 183 | 0 | 0
  Week 28 | 29.5 |  |
  Week 32: number analyzed (Participants) | 178 | 0 | 0
  Week 32 | 31.5 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 380
  Week 36 | 32.0 | 58.3 | 64.7
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 30.4 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 38.7 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 40.5 | 58.4 | 65.9
  Week 60: number analyzed (Participants) | 157 | 191 | 355
  Week 60 | 40.1 | 57.6 | 67.3
  Week 72: number analyzed (Participants) | 150 | 182 | 349
  Week 72 | 43.3 | 59.9 | 69.9
  Week 84: number analyzed (Participants) | 139 | 178 | 338
  Week 84 | 43.9 | 57.9 | 69.8
  Week 96: number analyzed (Participants) | 136 | 172 | 306
  Week 96 | 53.7 | 56.4 | 71.2
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 51.9 | 64.0 | 70.8
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 48.5 | 66.2 | 71.4
  Week 132: number analyzed (Participants) | 126 | 115 | 175
  Week 132 | 55.6 | 67.0 | 72.6
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 58.3 | 63.9 | 71.1
  Week 156: number analyzed (Participants) | 119 | 70 | 105
  Week 156 | 55.5 | 67.1 | 67.6
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 56.0 | 64.9 | 69.7
  Week 180: number analyzed (Participants) | 113 | 21 | 45
  Week 180 | 57.5 | 57.1 | 75.6
  Week 192: number analyzed (Participants) | 110 | 8 | 22
  Week 192 | 55.5 | 62.5 | 68.2
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 60.7 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 103 | 0 | 0
  Week 216 | 54.4 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 59.2 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 60.0 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 60.0 |  |
  Week 264: number analyzed (Participants) | 89 | 0 | 0
  Week 264 | 56.2 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 62.8 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 57.1 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 60.5 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 57.0 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 60.9 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 52.8 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 52.5 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 50.0 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT | 42.8 | 54.5 | 67.5
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 23.8 | 35.4 | 40.4

14. Secondary Outcome: Change From Baseline of Preceding Study in Tender Joint Count (TJC) (68 Joints) Through Week 372
Description: The participants were examined for the tender joints and the location was confirmed by the investigator who assessed the following 68 joints which included temporomandibular joints (2), sternoclavicular joints (2), acromioclavicular joints (2), shoulder joints (2), elbow joints (2), wrist joints (2), distal interphalangeal joints (8), proximal interphalangeal joints of both hands (10), metacarpophalangeal joints (10), hip joints (2), knee joints (2), ankle joints (2), tarsal bones (2), metatarsophalangeal joints (10), interphalangeal joint joints of toes (2), proximal interphalangeal joints of both feet (8). Higher TJC indicated greater disease activity.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
tender joint count
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | -4.3 (8.2) | -11.7 (8.8) | -11.5 (8.4)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -5.3 (7.9) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -5.7 (8.6) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -7.7 (8.8) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | -8.7 (8.5) | -11.8 (8.9) | -11.8 (8.1)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -9.4 (8.3) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -9.5 (8.4) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | -9.8 (9.0) | -11.9 (8.8) | -12.1 (8.0)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -10.0 (8.7) |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | -9.5 (8.2) |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | -10.0 (8.0) | -12.4 (8.8) | -12.3 (7.9)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -10.4 (8.1) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -10.9 (8.2) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | -10.7 (8.3) | -11.9 (8.8) | -12.3 (8.2)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -10.8 (8.3) | -11.9 (9.2) | -12.4 (8.3)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -10.4 (8.8) | -11.9 (9.4) | -12.8 (8.5)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -10.7 (8.7) | -11.9 (9.0) | -12.9 (8.3)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -10.8 (7.9) | -12.3 (9.5) | -13.1 (8.4)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -10.7 (8.2) | -12.3 (9.3) | -13.8 (8.9)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -10.6 (8.4) | -12.7 (9.5) | -13.5 (9.2)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -10.8 (8.3) | -12.8 (9.9) | -13.8 (9.0)
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | -11.1 (9.0) | -12.9 (9.5) | -13.3 (9.3)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -11.2 (8.4) | -14.1 (10.4) | -13.3 (9.7)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -11.3 (8.7) | -11.8 (10.0) | -13.2 (9.1)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -11.3 (8.5) | -12.2 (7.5) | -14.2 (9.9)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -11.4 (8.7) | -11.8 (5.6) | -13.2 (10.8)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -11.8 (7.8) | -8.0 (NA) — SD not estimable as there is only one participant. | -17.0 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -11.7 (8.1) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -11.7 (7.9) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -11.7 (8.0) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -11.8 (8.3) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -11.7 (8.4) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -12.0 (8.4) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -11.5 (8.5) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -11.5 (8.6) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -11.9 (8.6) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -12.0 (8.2) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -11.5 (6.6) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -11.2 (5.8) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -13.8 (5.6) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -23.0 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 223 | 412
  EOT | -10.2 (9.6) | -11.5 (9.4) | -12.6 (8.6)
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | -8.6 (9.8) | -9.1 (7.6) | -9.4 (9.9)

15. Secondary Outcome: Change From Baseline of Preceding Study in Swollen Joint Count (SJC) (66 Joints) Through Week 372
Description: The participants were examined for the swollen joints and the location was confirmed by the investigator who assessed the following 66 joints which included temporomandibular joints (2), sternoclavicular joints (2), acromioclavicular joints (2), shoulder joints (2), elbow joints (2), wrist joints (2), distal interphalangeal joints (8), proximal interphalangeal joints of both hands (10), metacarpophalangeal joints (10), knee joints (2), ankle joints (2), tarsal bones (2), metatarsophalangeal joints (10), interphalangeal joint joints of toes (2), proximal interphalangeal joints of both feet (8). Higher SJC indicated greater disease activity.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
swollen joint count
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | -3.8 (5.5) | -9.6 (6.9) | -10.5 (6.4)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -4.6 (5.8) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -4.8 (6.2) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -6.1 (6.3) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | -6.7 (6.1) | -9.5 (6.6) | -10.4 (6.4)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -7.1 (5.8) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -7.4 (6.1) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | -7.6 (5.9) | -9.9 (6.4) | -10.8 (6.4)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -7.6 (6.0) |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | -7.5 (5.7) |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | -7.9 (5.5) | -10.3 (6.6) | -11.1 (6.5)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -8.1 (5.5) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -8.6 (5.4) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | -8.7 (5.6) | -10.4 (6.4) | -11.0 (6.7)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -8.4 (6.1) | -10.3 (6.8) | -11.1 (6.6)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -8.6 (5.8) | -10.3 (6.6) | -11.3 (6.7)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -8.7 (5.6) | -10.2 (6.7) | -11.2 (6.6)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -8.8 (5.2) | -10.6 (7.0) | -11.3 (6.5)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -9.0 (5.3) | -10.7 (7.5) | -11.5 (6.9)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -8.7 (5.8) | -11.1 (7.3) | -11.4 (6.6)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -9.0 (5.7) | -11.2 (7.3) | -11.5 (6.8)
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | -9.1 (5.6) | -11.2 (7.8) | -11.3 (6.7)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -8.9 (5.7) | -12.4 (8.1) | -11.4 (7.0)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -9.2 (5.9) | -11.4 (7.0) | -11.7 (6.8)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -9.2 (5.4) | -10.6 (6.2) | -11.9 (7.3)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -9.1 (5.7) | -9.0 (7.3) | -11.3 (7.5)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -9.5 (5.5) | -6.0 (NA) — SD not estimable as there is only one participant. | -17.0 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -9.2 (6.0) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -9.4 (5.4) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -9.7 (5.8) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -9.6 (5.7) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -9.7 (5.5) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -9.9 (5.5) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -9.5 (5.7) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -9.7 (5.7) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -9.4 (5.8) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -9.5 (5.7) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -9.4 (5.3) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -9.4 (5.1) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -11.0 (5.8) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -18.0 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 223 | 412
  EOT | -7.8 (6.6) | -9.7 (7.1) | -11.1 (6.8)
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | -6.3 (7.2) | -8.2 (7.4) | -9.3 (7.6)

16. Secondary Outcome: Change From Baseline of Preceding Study in CRP (mg/dL) Through Week 372
Description: Higher CRP indicates greater disease activity.
Time Frame: Baseline of preceding study and weeks 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144,156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, 312, 324, 336, 348, 360, 372, EOT, EOS
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
mg/dL
  Week 0: number analyzed (Participants) | 200 | 224 | 411
  Week 0 | -0.334 (1.691) | -1.590 (2.106) | -1.932 (2.014)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -0.752 (1.724) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -0.745 (1.897) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -1.032 (1.932) |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | -1.034 (2.225) | -1.528 (2.121) | -1.932 (2.037)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -1.176 (2.203) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -1.242 (2.221) |  |
  Week 24: number analyzed (Participants) | 187 | 208 | 394
  Week 24 | -1.237 (2.168) | -1.507 (2.129) | -1.991 (2.125)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -1.376 (2.039) |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | -1.296 (2.040) |  |
  Week 36: number analyzed (Participants) | 172 | 207 | 381
  Week 36 | -1.330 (2.073) | -1.552 (2.087) | -2.031 (2.116)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -1.361 (2.217) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -1.361 (2.260) |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | -1.367 (2.070) | -1.604 (2.096) | -2.088 (2.034)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -1.310 (2.011) | -1.534 (2.163) | -2.063 (2.062)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -1.456 (2.165) | -1.726 (2.008) | -2.019 (2.023)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -1.418 (2.159) | -1.501 (2.337) | -1.991 (2.092)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -1.485 (2.113) | -1.561 (2.101) | -1.983 (2.606)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -1.562 (2.060) | -1.565 (2.444) | -2.066 (1.990)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -1.507 (2.199) | -1.730 (2.163) | -1.964 (2.108)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -1.443 (2.602) | -1.519 (2.231) | -2.058 (2.178)
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | -1.609 (2.297) | -1.474 (2.155) | -2.120 (2.329)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -1.423 (2.489) | -1.731 (1.892) | -2.432 (2.277)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -1.576 (2.213) | -1.418 (2.153) | -2.211 (2.227)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -1.170 (2.340) | -2.088 (1.984) | -2.230 (2.053)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -1.506 (1.976) | -1.501 (1.575) | -2.060 (2.014)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -1.477 (2.154) | -1.570 (NA) — SD not estimable as there is only one participant. | -0.950 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -1.374 (2.209) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -1.449 (2.232) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -1.440 (2.340) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -1.488 (2.263) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -1.498 (2.379) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -1.647 (2.264) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -1.580 (2.404) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -1.537 (2.470) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -1.263 (2.319) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -1.565 (2.238) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -1.452 (2.189) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -1.365 (2.015) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -2.179 (2.117) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -2.330 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | -1.072 (2.470) | -1.386 (2.340) | -1.845 (2.438)
  EOS: number analyzed (Participants) | 101 | 66 | 89
  EOS | -0.967 (2.251) | -1.262 (2.930) | -1.270 (2.818)

17. Secondary Outcome: Change From Baseline of Preceding Study in ESR (mm/h) Through Week 372
Description: Higher ESR indicates greater disease activity.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
mm/h
  Week 0: number analyzed (Participants) | 200 | 223 | 410
  Week 0 | -2.46 (17.83) | -22.66 (25.31) | -27.02 (23.11)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -6.65 (18.03) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -6.93 (18.01) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -10.54 (17.93) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 407
  Week 12 | -11.93 (18.44) | -22.43 (26.18) | -27.72 (23.47)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -13.39 (19.30) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -14.07 (17.92) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 392
  Week 24 | -14.45 (18.12) | -22.91 (25.13) | -28.54 (24.45)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -15.15 (17.28) |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | -16.20 (17.74) |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 380
  Week 36 | -16.26 (19.70) | -22.51 (26.62) | -29.41 (23.34)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -16.27 (19.89) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -15.60 (20.47) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 366
  Week 48 | -16.09 (19.14) | -23.63 (25.51) | -30.31 (23.67)
  Week 60: number analyzed (Participants) | 157 | 190 | 355
  Week 60 | -16.71 (19.07) | -23.34 (24.86) | -30.06 (23.69)
  Week 72: number analyzed (Participants) | 150 | 182 | 348
  Week 72 | -16.78 (21.18) | -24.70 (24.16) | -30.06 (23.85)
  Week 84: number analyzed (Participants) | 140 | 178 | 337
  Week 84 | -16.89 (20.87) | -22.58 (26.95) | -29.23 (24.23)
  Week 96: number analyzed (Participants) | 136 | 172 | 306
  Week 96 | -18.81 (21.28) | -21.71 (25.55) | -29.70 (25.14)
  Week 108: number analyzed (Participants) | 133 | 163 | 266
  Week 108 | -19.24 (20.02) | -22.46 (25.87) | -29.97 (25.60)
  Week 120: number analyzed (Participants) | 130 | 147 | 212
  Week 120 | -19.48 (21.41) | -24.36 (25.63) | -29.46 (25.87)
  Week 132: number analyzed (Participants) | 126 | 115 | 175
  Week 132 | -19.43 (23.78) | -22.13 (26.42) | -30.35 (24.34)
  Week 144: number analyzed (Participants) | 120 | 96 | 135
  Week 144 | -22.19 (22.29) | -21.48 (22.87) | -31.44 (24.17)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -20.62 (23.11) | -23.14 (23.91) | -30.77 (25.02)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -20.58 (22.98) | -24.95 (22.89) | -29.68 (22.86)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -16.28 (23.48) | -23.52 (28.44) | -33.46 (24.70)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -18.86 (20.85) | -38.63 (35.76) | -26.50 (27.72)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -19.05 (21.63) | -11.00 (NA) — SD not estimable as there is only one participant. | -57.00 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -17.85 (23.11) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -20.09 (22.96) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -19.24 (22.01) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -20.78 (21.72) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -19.11 (24.20) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -20.21 (21.14) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -17.57 (25.36) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -19.51 (20.15) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -16.81 (21.06) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -17.28 (22.08) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -17.51 (21.38) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -16.53 (21.63) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -20.63 (22.81) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -28.00 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 223 | 411
  EOT | -12.52 (21.92) | -20.04 (26.47) | -26.36 (27.00)
  EOS: number analyzed (Participants) | 101 | 66 | 89
  EOS | -8.90 (24.70) | -14.48 (25.73) | -17.26 (27.20)

18. Secondary Outcome: Percentage of Participants Achieving ACR/European League Against Rheumatism (EULAR) Response Through Week 372
Description: ACR/EULAR Remission was defined as TJC (68 joints) ≤ 1, SJC (66 joints) ≤1, CRP ≤1 mg/dL, and participant's global assessment of arthritis ≤ 1 cm (on a visual analog scale (VAS) of 0 - 100 mm).
Time Frame: as for outcome 10
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 224 | 411
  Week 0 | 1.5 | 18.3 | 22.4
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 4.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 5.0 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 4.5 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 4.0 | 16.9 | 23.0
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 7.1 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 7.4 |  |
  Week 24: number analyzed (Participants) | 187 | 208 | 394
  Week 24 | 7.5 | 20.2 | 26.9
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 9.2 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 10.6 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 381
  Week 36 | 11.0 | 29.1 | 28.3
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 8.3 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 11.0 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 11.0 | 25.9 | 32.7
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 10.8 | 24.1 | 28.9
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 11.3 | 29.5 | 30.7
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 14.3 | 30.0 | 34.0
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 17.5 | 26.6 | 33.2
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 18.0 | 28.7 | 30.0
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 16.9 | 29.1 | 26.3
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 20.6 | 29.3 | 31.4
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 18.3 | 30.9 | 28.9
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 17.6 | 27.1 | 31.1
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 21.6 | 35.1 | 31.6
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 21.1 | 23.8 | 34.8
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 21.6 | 25.0 | 31.8
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 23.4 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 25.0 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 24.5 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 24.2 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 25.6 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 24.4 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 19.8 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 25.0 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 24.7 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 24.1 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 23.4 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 24.5 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 15.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 25.0 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0.0 |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | 15.9 | 25.7 | 31.3
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 10.9 | 7.7 | 12.4

19. Secondary Outcome: Percentage of Participants With a EULAR Good Response Using DAS28-CRP Through Week 372
Description: The Disease Activity Score Based on 28-joints Count based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to =<5.1 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1. Percentage of participants with good response have been reported in this outcome measure.
Time Frame: as for outcome 2
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 224 | 411
  Week 0 | 11.5 | 71.0 | 71.0
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 18.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 19.6 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 27.1 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 34.8 | 70.3 | 72.3
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 36.2 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 43.7 |  |
  Week 24: number analyzed (Participants) | 187 | 208 | 394
  Week 24 | 44.4 | 70.2 | 77.2
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 47.8 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 46.4 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 381
  Week 36 | 49.4 | 72.3 | 78.2
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 53.0 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 53.4 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 56.4 | 73.1 | 80.1
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 58.0 | 71.7 | 82.3
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 59.3 | 76.5 | 84.0
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 63.6 | 75.0 | 82.0
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 72.3 | 77.5 | 84.0
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 72.9 | 75.6 | 85.8
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 70.8 | 83.8 | 85.4
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 73.8 | 80.2 | 85.7
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 78.3 | 80.4 | 85.2
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 74.8 | 75.7 | 84.9
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 73.3 | 75.7 | 86.8
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 71.9 | 76.2 | 84.8
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 74.8 | 87.5 | 86.4
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 77.6 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 73.1 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 79.6 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 78.9 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 76.7 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 80.0 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 81.4 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 78.6 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 80.2 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 81.0 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 79.7 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 71.7 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 75.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 100.0 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | 58.7 | 69.4 | 83.3
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 38.6 | 43.1 | 58.4

20. Secondary Outcome: Percentage of Participants With a EULAR Good Response Using DAS28-ESR Through Week 372
Description: The Disease Activity Score Based on 28-joints Count based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to =<5.1 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1. Percentage of participants with good response have been reported in the outcome measure.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 411
  Week 0 | 7.0 | 54.7 | 54.5
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 11.5 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 13.1 |  |
  Week 8: number analyzed (Participants) | 197 | 0 | 0
  Week 8 | 13.7 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 21.7 | 50.7 | 58.1
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 21.9 |  |
  Week 20: number analyzed (Participants) | 189 | 0 | 0
  Week 20 | 23.3 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 393
  Week 24 | 27.3 | 52.7 | 61.6
  Week 28: number analyzed (Participants) | 183 | 0 | 0
  Week 28 | 29.0 |  |
  Week 32: number analyzed (Participants) | 178 | 0 | 0
  Week 32 | 30.9 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 380
  Week 36 | 30.8 | 54.9 | 63.7
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 28.6 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 36.8 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 38.0 | 56.3 | 65.1
  Week 60: number analyzed (Participants) | 157 | 191 | 355
  Week 60 | 39.5 | 55.5 | 66.5
  Week 72: number analyzed (Participants) | 150 | 182 | 349
  Week 72 | 42.7 | 58.2 | 68.5
  Week 84: number analyzed (Participants) | 139 | 178 | 338
  Week 84 | 43.9 | 54.5 | 68.6
  Week 96: number analyzed (Participants) | 136 | 172 | 306
  Week 96 | 51.5 | 54.7 | 69.6
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 50.4 | 61.6 | 68.9
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 46.2 | 64.2 | 69.5
  Week 132: number analyzed (Participants) | 126 | 115 | 175
  Week 132 | 54.0 | 64.3 | 71.4
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 56.7 | 60.8 | 68.9
  Week 156: number analyzed (Participants) | 119 | 70 | 105
  Week 156 | 53.8 | 65.7 | 67.6
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 55.2 | 64.9 | 68.4
  Week 180: number analyzed (Participants) | 113 | 21 | 45
  Week 180 | 56.6 | 57.1 | 73.3
  Week 192: number analyzed (Participants) | 110 | 8 | 22
  Week 192 | 54.5 | 62.5 | 63.6
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 59.8 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 103 | 0 | 0
  Week 216 | 52.4 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 58.2 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 56.8 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 57.8 |  |
  Week 264: number analyzed (Participants) | 89 | 0 | 0
  Week 264 | 56.2 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 60.5 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 54.8 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 58.0 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 54.4 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 59.4 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 50.9 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 52.5 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 50.0 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT | 41.3 | 52.2 | 65.8
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 20.8 | 35.4 | 40.4

21. Secondary Outcome: Percentage of Participants With a EULAR Good or Moderate Response Using DAS28-ESR Through Week 372
Description: The Disease Activity Score Based on 28-joints Count based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to =<5.1 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1. Percentage of participants with good or moderate response have been reported in this outcome measure.
Time Frame: as for outcome 2
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 411
  Week 0 | 41.5 | 89.7 | 93.4
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 54.5 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 59.3 |  |
  Week 8: number analyzed (Participants) | 197 | 0 | 0
  Week 8 | 70.1 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 75.8 | 91.3 | 92.2
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 78.1 |  |
  Week 20: number analyzed (Participants) | 189 | 0 | 0
  Week 20 | 85.2 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 393
  Week 24 | 84.0 | 92.3 | 95.4
  Week 28: number analyzed (Participants) | 183 | 0 | 0
  Week 28 | 87.4 |  |
  Week 32: number analyzed (Participants) | 178 | 0 | 0
  Week 32 | 84.8 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 380
  Week 36 | 91.3 | 92.2 | 95.5
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 89.3 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 93.3 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 92.6 | 94.4 | 95.1
  Week 60: number analyzed (Participants) | 157 | 191 | 355
  Week 60 | 93.0 | 92.1 | 94.9
  Week 72: number analyzed (Participants) | 150 | 182 | 349
  Week 72 | 90.7 | 91.2 | 96.0
  Week 84: number analyzed (Participants) | 139 | 178 | 338
  Week 84 | 89.9 | 92.7 | 95.9
  Week 96: number analyzed (Participants) | 136 | 172 | 306
  Week 96 | 92.6 | 94.2 | 97.1
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 92.5 | 91.5 | 97.4
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 91.5 | 93.9 | 96.2
  Week 132: number analyzed (Participants) | 126 | 115 | 175
  Week 132 | 92.1 | 89.6 | 97.7
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 93.3 | 87.6 | 97.0
  Week 156: number analyzed (Participants) | 119 | 70 | 105
  Week 156 | 94.1 | 95.7 | 96.2
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 92.2 | 86.5 | 96.1
  Week 180: number analyzed (Participants) | 113 | 21 | 45
  Week 180 | 93.8 | 90.5 | 93.3
  Week 192: number analyzed (Participants) | 110 | 8 | 22
  Week 192 | 94.5 | 87.5 | 95.5
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 95.3 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 103 | 0 | 0
  Week 216 | 93.2 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 92.9 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 92.6 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 92.2 |  |
  Week 264: number analyzed (Participants) | 89 | 0 | 0
  Week 264 | 92.1 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 94.2 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 92.9 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 95.1 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 94.9 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 96.9 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 94.3 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 92.5 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 100.0 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT | 76.6 | 87.1 | 93.7
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 67.3 | 80.0 | 82.0

22. Secondary Outcome: Percentage of Participants With a EULAR Good or Moderate Response Using DAS28-CRP Through Week 372
Description: as for outcome 21
Time Frame: as for outcome 2
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 224 | 411
  Week 0 | 48.5 | 94.2 | 94.6
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 60.5 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 65.8 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 75.4 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 79.8 | 92.7 | 94.9
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 81.6 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 84.2 |  |
  Week 24: number analyzed (Participants) | 187 | 208 | 394
  Week 24 | 84.5 | 95.2 | 96.2
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 88.0 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 88.3 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 381
  Week 36 | 91.3 | 95.1 | 96.9
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 92.9 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 93.3 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 92.0 | 94.9 | 97.3
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 94.9 | 93.7 | 96.1
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 92.7 | 95.1 | 96.3
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 92.1 | 95.0 | 96.4
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 94.2 | 94.2 | 97.7
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 95.5 | 93.9 | 98.1
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 93.1 | 98.0 | 96.7
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 92.1 | 94.0 | 97.7
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 95.0 | 90.7 | 96.3
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 94.1 | 97.1 | 98.1
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 94.0 | 94.6 | 98.7
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 93.9 | 95.2 | 97.8
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 95.5 | 87.5 | 95.5
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 96.3 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 94.2 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 93.9 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 94.7 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 93.3 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 91.1 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 95.3 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 94.0 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 93.8 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 94.9 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 98.4 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 98.1 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 92.5 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 100.0 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | 78.6 | 89.2 | 95.4
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 72.3 | 80.0 | 83.1

23. Secondary Outcome: Percentage of Participants With a Simplified Disease Activity Index (SDAI) Score of <= 3.3 Through Week 372
Description: SDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, CRP (mg/dL), and calculated according to description. SDAI = TJC + SJC + SGA + PGA + CRP. The SDAI score ranges from 0 to approximately 86. Higher SDAI indicates greater disease activity. SDAI Remission was defined as SDAI score ≤ 3.3.
Time Frame: as for outcome 10
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 224 | 411
  Week 0 | 4.0 | 24.6 | 32.6
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 5.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 6.0 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 5.5 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 6.1 | 27.4 | 31.4
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 8.7 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 10.0 |  |
  Week 24: number analyzed (Participants) | 187 | 208 | 394
  Week 24 | 13.4 | 28.4 | 37.1
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 15.2 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 16.2 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 381
  Week 36 | 16.9 | 31.6 | 40.9
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 12.5 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 16.6 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 18.4 | 32.5 | 42.8
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 14.0 | 30.4 | 41.6
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 21.3 | 37.7 | 43.3
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 21.4 | 35.6 | 42.3
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 24.1 | 37.6 | 42.0
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 25.6 | 39.6 | 42.7
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 24.6 | 40.5 | 38.0
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 28.6 | 41.4 | 44.0
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | 27.5 | 41.2 | 45.2
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 24.4 | 42.9 | 42.5
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 28.4 | 51.4 | 44.7
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 27.2 | 42.9 | 45.7
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 33.3 | 25.0 | 50.0
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 30.8 | 0.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 33.7 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 37.8 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 37.9 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 31.1 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 35.6 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 32.6 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 38.1 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 33.3 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 32.9 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 34.4 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 28.3 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 22.5 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 31.3 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0.0 |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | 23.9 | 36.0 | 43.4
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 13.9 | 13.8 | 24.7

24. Secondary Outcome: Change From Baseline of Preceding Study in SDAI Score Through Week 372
Description: SDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, CRP (mg/dL), and calculated according to description: SDAI = TJC + SJC + SGA + PGA + CRP. The SDAI score ranges from 0 to approximately 86. Higher SDAI indicates greater disease activity.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 411
  Week 0 | -7.41 (11.53) | -24.30 (13.03) | -25.12 (12.32)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -10.13 (11.06) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -10.93 (12.01) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -14.33 (12.03) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | -16.14 (12.02) | -23.93 (13.02) | -25.15 (12.17)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -17.53 (11.95) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -18.11 (12.16) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | -18.61 (11.99) | -24.13 (12.84) | -25.93 (11.90)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -19.43 (12.07) |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | -18.66 (12.25) |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | -19.62 (11.23) | -25.00 (13.12) | -26.45 (11.70)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -20.26 (11.40) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -20.96 (11.46) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | -21.17 (11.97) | -24.93 (12.56) | -26.75 (11.98)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -21.10 (12.21) | -24.54 (13.27) | -26.73 (12.04)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -21.65 (13.09) | -25.17 (13.02) | -27.31 (12.04)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -21.82 (12.90) | -24.70 (13.34) | -27.15 (12.02)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -22.40 (12.25) | -25.37 (13.36) | -27.52 (11.72)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -22.73 (12.74) | -25.38 (13.68) | -28.28 (12.38)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -22.18 (13.61) | -26.57 (13.40) | -27.71 (12.37)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -22.90 (13.51) | -26.38 (14.24) | -27.83 (12.16)
  Week 144: number analyzed (Participants) | 120 | 97 | 135
  Week 144 | -23.58 (12.96) | -26.53 (14.75) | -27.38 (13.05)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -23.19 (13.04) | -28.68 (15.05) | -28.07 (13.27)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -23.64 (13.12) | -26.75 (15.71) | -27.34 (13.31)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -23.07 (13.37) | -26.63 (15.13) | -29.04 (13.67)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -23.75 (13.34) | -24.37 (15.48) | -27.99 (13.04)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -24.42 (12.08) | -26.92 (NA) — SD not estimable as there is only one participant. | -36.00 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -24.00 (12.81) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -24.18 (12.64) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -24.55 (12.88) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -24.47 (13.18) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -24.36 (13.22) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -25.23 (12.77) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -24.71 (13.15) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -24.56 (13.46) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -24.52 (13.38) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -25.45 (12.83) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -23.68 (12.34) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -22.45 (11.80) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -27.23 (11.15) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -53.18 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 221 | 412
  EOT | -19.12 (15.01) | -23.68 (14.37) | -26.58 (13.07)
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | -14.81 (13.90) | -19.25 (14.64) | -20.05 (14.05)

25. Secondary Outcome: Percentage of Participants With a Clinical Disease Activity Index (CDAI) Score of <= 2.8 Through Week 372
Description: CDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA (0-10 cm VAS), PGA (0-10 cm VAS), and calculated according to description: CDAI = TJC + SJC + SGA + PGA. The CDAI score ranges from 0 to approximately 76. CDAI. Remission was defined as CDAI score ≤ 2.8.
Time Frame: as for outcome 2
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 224 | 412
  Week 0 | 3.0 | 23.7 | 30.6
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 4.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 4.5 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 6.0 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 5.6 | 24.2 | 30.6
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 7.7 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 8.9 |  |
  Week 24: number analyzed (Participants) | 187 | 208 | 394
  Week 24 | 11.8 | 29.3 | 36.0
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 14.1 |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | 16.8 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 381
  Week 36 | 15.1 | 30.6 | 39.1
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 13.7 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 15.3 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 19.6 | 33.5 | 42.2
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 14.0 | 28.3 | 40.7
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 18.7 | 36.6 | 42.4
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 20.0 | 33.9 | 42.6
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 23.4 | 37.6 | 42.7
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 26.3 | 37.2 | 40.4
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 23.1 | 39.9 | 39.0
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 25.4 | 44.0 | 42.3
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 25.0 | 42.3 | 44.9
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 19.3 | 41.4 | 40.6
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 28.4 | 51.4 | 43.4
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 28.1 | 33.3 | 43.5
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 30.6 | 25.0 | 45.5
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 29.9 | 0.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 33.7 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 33.7 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 34.7 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 30.0 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 31.1 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 31.4 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 38.1 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 30.9 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 31.6 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 34.4 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 26.4 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 20.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 31.3 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0.0 |  |
  EOT: number analyzed (Participants) | 201 | 223 | 412
  EOT | 24.9 | 34.5 | 42.5
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 14.9 | 12.3 | 25.8

26. Secondary Outcome: Change From Baseline of Preceding Study CDAI Score Through Week 372
Description: CDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA (0-10 cm VAS), PGA (0-10 cm VAS), and calculated according to description: CDAI = TJC + SJC + SGA + PGA. The CDAI score ranges from 0 to approximately 76. Higher CDAI indicates greater disease activity.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | -7.07 (10.78) | -22.70 (12.24) | -23.22 (11.73)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -9.38 (10.44) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -10.19 (11.36) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -13.30 (11.28) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | -15.11 (11.10) | -22.39 (12.28) | -23.21 (11.54)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -16.35 (10.88) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -16.87 (11.15) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | -17.37 (11.35) | -22.62 (12.17) | -23.93 (11.24)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -18.06 (11.39) |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | -17.36 (11.37) |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | -18.29 (10.42) | -23.41 (12.39) | -24.42 (11.13)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -18.90 (10.50) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -19.60 (10.58) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | -19.80 (11.03) | -23.32 (11.98) | -24.66 (11.45)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -19.79 (11.41) | -23.01 (12.53) | -24.66 (11.53)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -20.19 (12.16) | -23.45 (12.39) | -25.29 (11.55)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -20.40 (12.11) | -23.20 (12.61) | -25.16 (11.54)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -20.92 (11.41) | -23.81 (12.62) | -25.54 (11.27)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -21.17 (11.87) | -23.81 (12.76) | -26.22 (11.82)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -20.68 (12.79) | -24.84 (12.73) | -25.74 (11.66)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -21.46 (12.30) | -24.86 (13.57) | -25.77 (11.56)
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | -21.97 (11.87) | -25.06 (14.11) | -25.23 (12.10)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -21.77 (11.89) | -26.95 (14.59) | -25.64 (12.50)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -22.06 (12.12) | -25.34 (14.99) | -25.13 (12.55)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -21.90 (12.27) | -24.54 (14.26) | -26.81 (13.07)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -22.24 (12.55) | -22.87 (14.41) | -25.93 (12.65)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -22.95 (11.32) | -25.35 (NA) — SD not estimable as there is only one participant. | -35.05 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -22.62 (11.84) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -22.73 (11.89) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -23.11 (11.88) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -22.98 (12.28) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -22.86 (12.21) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -23.58 (11.91) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -23.13 (12.18) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -23.02 (12.27) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -23.26 (12.34) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -23.89 (11.85) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -22.23 (11.56) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -21.08 (11.11) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -25.05 (10.77) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -50.85 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | -18.05 (13.98) | -22.24 (13.54) | -24.74 (12.26)
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | -13.84 (13.08) | -17.97 (12.75) | -18.78 (12.87)

27. Secondary Outcome: Change From Baseline of Preceding Study in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score Through Week 108
Description: FACIT-Fatigue was used to assess the burden of self-reported fatigue caused by a chronic disease and its impact upon daily activities and function. It has 13-items with symptom-specific questions, each of the 13 items of the FACIT-Fatigue scale ranges from 0 (Not at all) - 4 (Very much), the range of possible scores is 0 - 52. Higher scores indicate higher fatigue.
Time Frame: Baseline of preceding study and weeks 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, EOT, EOS
Population: FAS population with available data at each time point. Only 015K-CL-RAJ1 arm was analyzed for this outcome as planned.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1
Number analyzed (Participants) | 201
units on a scale
  Week 0: number analyzed (Participants) | 200
  Week 0 | 1.71 (8.52)
  Week 2: number analyzed (Participants) | 2
  Week 2 | 4.50 (3.54)
  Week 4: number analyzed (Participants) | 199
  Week 4 | 3.29 (8.08)
  Week 8: number analyzed (Participants) | 199
  Week 8 | 4.15 (8.66)
  Week 12: number analyzed (Participants) | 198
  Week 12 | 4.85 (8.79)
  Week 16: number analyzed (Participants) | 196
  Week 16 | 5.91 (8.50)
  Week 20: number analyzed (Participants) | 190
  Week 20 | 5.86 (9.26)
  Week 24: number analyzed (Participants) | 187
  Week 24 | 5.99 (8.93)
  Week 28: number analyzed (Participants) | 184
  Week 28 | 5.95 (8.96)
  Week 32: number analyzed (Participants) | 180
  Week 32 | 5.91 (8.49)
  Week 36: number analyzed (Participants) | 172
  Week 36 | 5.91 (8.72)
  Week 40: number analyzed (Participants) | 168
  Week 40 | 6.06 (8.87)
  Week 44: number analyzed (Participants) | 163
  Week 44 | 6.05 (8.40)
  Week 48: number analyzed (Participants) | 163
  Week 48 | 6.34 (8.44)
  Week 60: number analyzed (Participants) | 138
  Week 60 | 7.18 (9.03)
  Week 72: number analyzed (Participants) | 113
  Week 72 | 5.87 (8.90)
  Week 84: number analyzed (Participants) | 76
  Week 84 | 6.11 (8.15)
  Week 96: number analyzed (Participants) | 39
  Week 96 | 6.10 (8.22)
  Week 108: number analyzed (Participants) | 1
  Week 108 | -6.0 (NA) — SD not estimable as data reported for one participant.
  EOT | 5.95 (9.24)
  EOS: number analyzed (Participants) | 6
  EOS | 3.67 (9.77)

28. Secondary Outcome: Change From Baseline of Preceding Study in Work Productivity and Activity Impairment Questionnaire (WPAI) Percent Work Time Missed Through Week 192
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work). Higher WPAI scores indicated greater activity impairment. The scores were multiplied by 100 to express in percentages. Percent work time missed due to problem was calculated as Q2/(Q2+Q4). Negative values indicate improvement from baseline.
Time Frame: Baseline of preceding study and weeks 0, 24, 48, 72, 96, 120, 144, 168, 192, EOT
Population: FAS population with available data at each time point. Only 015K-CL-RAJ3 and 015K-CL-RAJ4 arms were analyzed for this outcome as planned.
Measure: Mean (Standard Deviation); unit: percent work time missed
Arm/Group | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 116 | 211
percent work time missed
  Week 0: number analyzed (Participants) | 116 | 210
  Week 0 | -5.36 (16.76) | -2.20 (18.46)
  Week 24: number analyzed (Participants) | 105 | 194
  Week 24 | -4.81 (17.40) | -3.29 (14.30)
  Week 48: number analyzed (Participants) | 102 | 181
  Week 48 | -4.52 (19.86) | -3.30 (17.16)
  Week 72: number analyzed (Participants) | 96 | 174
  Week 72 | -4.73 (18.43) | -3.17 (15.47)
  Week 96: number analyzed (Participants) | 93 | 151
  Week 96 | -4.74 (19.00) | -3.13 (14.38)
  Week 120: number analyzed (Participants) | 77 | 103
  Week 120 | -5.15 (20.38) | -4.49 (17.14)
  Week 144: number analyzed (Participants) | 53 | 68
  Week 144 | -3.21 (14.26) | -1.26 (20.09)
  Week 168: number analyzed (Participants) | 17 | 35
  Week 168 | -8.65 (21.30) | -5.19 (19.82)
  Week 192: number analyzed (Participants) | 2 | 10
  Week 192 | 0.00 (0.00) | -2.29 (6.62)
  EOT | -2.76 (20.13) | -1.96 (17.64)

29. Secondary Outcome: Change From Baseline of Preceding Study in WPAI Percent Impairment While Working Through Week 192
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work). Higher WPAI scores indicated greater activity impairment. The scores were multiplied by 100 to express in percentages. Percent impairment while working due to problem was calculated as Q5/10. Negative values indicate improvement from baseline.
Time Frame: Baseline of preceding study and weeks 0, 24, 48, 72, 96, 120, 144, 168, 192, EOT
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: percent work impairment
Arm/Group | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 114 | 208
percent work impairment
  Week 0: number analyzed (Participants) | 114 | 206
  Week 0 | -21.05 (33.06) | -22.18 (28.64)
  Week 24: number analyzed (Participants) | 103 | 192
  Week 24 | -21.94 (32.60) | -24.79 (26.64)
  Week 48: number analyzed (Participants) | 100 | 178
  Week 48 | -20.70 (31.82) | -25.17 (27.33)
  Week 72: number analyzed (Participants) | 94 | 170
  Week 72 | -21.06 (31.47) | -27.12 (27.72)
  Week 96: number analyzed (Participants) | 91 | 151
  Week 96 | -20.11 (31.39) | -28.54 (26.94)
  Week 120: number analyzed (Participants) | 75 | 102
  Week 120 | -24.40 (30.15) | -30.00 (29.38)
  Week 144: number analyzed (Participants) | 52 | 67
  Week 144 | -18.08 (30.62) | -27.16 (31.37)
  Week 168: number analyzed (Participants) | 17 | 34
  Week 168 | -17.06 (34.96) | -23.24 (31.79)
  Week 192: number analyzed (Participants) | 2 | 10
  Week 192 | -15.00 (21.21) | -28.00 (35.53)
  EOT | -21.49 (33.56) | -24.13 (29.46)

30. Secondary Outcome: Change From Baseline of Preceding Study in WPAI Percent Overall Work Impairment Through Week 192
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work). Higher WPAI scores indicated greater activity impairment. The scores were multiplied by 100 to express in percentages. Percent overall work impairment due to problem was calculated as Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)]. Negative values indicate improvement from baseline.
Time Frame: Baseline of preceding study and weeks 0, 24, 48, 72, 96, 120, 144, 168, 192, EOT
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: percent overall work impairment
Arm/Group | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 114 | 208
percent overall work impairment
  Week 0: number analyzed (Participants) | 114 | 206
  Week 0 | -22.24 (33.23) | -22.20 (30.83)
  Week 24: number analyzed (Participants) | 103 | 192
  Week 24 | -22.45 (32.86) | -25.78 (27.99)
  Week 48: number analyzed (Participants) | 100 | 178
  Week 48 | -20.80 (32.72) | -25.32 (30.00)
  Week 72: number analyzed (Participants) | 94 | 170
  Week 72 | -21.59 (32.40) | -27.41 (28.98)
  Week 96: number analyzed (Participants) | 91 | 150
  Week 96 | -20.58 (32.29) | -28.93 (28.34)
  Week 120: number analyzed (Participants) | 75 | 101
  Week 120 | -24.71 (30.92) | -31.40 (30.13)
  Week 144: number analyzed (Participants) | 52 | 67
  Week 144 | -18.29 (31.64) | -26.76 (33.82)
  Week 168: number analyzed (Participants) | 17 | 34
  Week 168 | -19.03 (36.72) | -24.76 (32.39)
  Week 192: number analyzed (Participants) | 2 | 10
  Week 192 | -15.00 (21.21) | -28.06 (36.25)
  EOT | -20.75 (33.46) | -24.63 (31.29)

31. Secondary Outcome: Change From Baseline of Preceding Study in WPAI Percent Activity Impairment Through Week 192
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicated greater activity impairment. The scores were multiplied by 100 to express in percentages. Percent activity impairment due to problem was calculated as Q6/10. Negative values indicate improvement from baseline.
Time Frame: Baseline of preceding study and weeks 0, 24, 48, 72, 96, 120, 144, 168, 192, EOT
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: percent activity impairment
Arm/Group | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 223 | 410
percent activity impairment
  Week 0 | -28.16 (29.69) | -25.39 (29.77)
  Week 24: number analyzed (Participants) | 206 | 392
  Week 24 | -27.38 (30.15) | -29.31 (28.92)
  Week 48: number analyzed (Participants) | 196 | 366
  Week 48 | -27.81 (30.76) | -28.85 (29.34)
  Week 72: number analyzed (Participants) | 183 | 347
  Week 72 | -28.09 (31.12) | -31.59 (30.71)
  Week 96: number analyzed (Participants) | 173 | 304
  Week 96 | -27.92 (30.69) | -30.69 (29.30)
  Week 120: number analyzed (Participants) | 148 | 212
  Week 120 | -29.26 (31.56) | -33.07 (30.69)
  Week 144: number analyzed (Participants) | 97 | 135
  Week 144 | -26.39 (32.57) | -31.11 (30.68)
  Week 168: number analyzed (Participants) | 37 | 75
  Week 168 | -20.81 (26.71) | -26.53 (31.64)
  Week 192: number analyzed (Participants) | 8 | 22
  Week 192 | -20.00 (30.24) | -23.18 (32.13)
  EOT: number analyzed (Participants) | 218 | 403
  EOT | -25.55 (32.04) | -27.87 (32.40)

32. Secondary Outcome: Percentage of Participants Achieving Health Assessment Questionnaire - Disability Index (HAQ-DI) Score <= 0.5 Through Week 372
Description: Participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item was scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: as for outcome 10
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 224 | 412
  Week 0 | 37.0 | 61.2 | 62.1
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 38.5 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 38.7 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 39.7 |  |
  Week 12: number analyzed (Participants) | 198 | 219 | 408
  Week 12 | 42.9 | 62.1 | 63.0
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 46.9 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 47.4 |  |
  Week 24: number analyzed (Participants) | 187 | 208 | 394
  Week 24 | 48.7 | 64.9 | 65.5
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 50.5 |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | 50.0 |  |
  Week 36: number analyzed (Participants) | 172 | 207 | 381
  Week 36 | 51.2 | 62.8 | 64.3
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 52.4 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 55.2 |  |
  Week 48: number analyzed (Participants) | 163 | 197 | 367
  Week 48 | 54.0 | 58.9 | 65.4
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 55.4 | 62.8 | 67.1
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 60.0 | 67.2 | 68.8
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 62.9 | 65.6 | 69.2
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 62.0 | 63.0 | 69.1
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 62.4 | 62.2 | 67.4
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 63.1 | 69.6 | 68.1
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 66.7 | 70.7 | 68.0
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 66.7 | 71.1 | 69.9
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 65.5 | 68.6 | 67.0
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 67.2 | 73.0 | 68.4
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 68.4 | 71.4 | 73.9
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 67.6 | 87.5 | 59.1
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 67.3 | 100.0 | 0.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 72.1 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 70.4 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 68.4 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 68.9 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 67.8 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 72.1 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 70.2 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 69.1 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 67.1 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 70.3 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 62.3 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 60.0 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 56.3 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT: number analyzed (Participants) | 201 | 223 | 412
  EOT | 52.7 | 62.3 | 63.6
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 35.6 | 40.0 | 48.3

33. Secondary Outcome: Change From Baseline of Preceding Study in HAQ-DI Through Week 372
Description: as for outcome 32
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | -0.03 (0.47) | -0.43 (0.57) | -0.49 (0.55)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -0.07 (0.44) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -0.08 (0.44) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -0.13 (0.47) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | -0.17 (0.45) | -0.44 (0.57) | -0.48 (0.59)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -0.21 (0.45) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -0.22 (0.46) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | -0.25 (0.46) | -0.43 (0.60) | -0.52 (0.59)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -0.27 (0.46) |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | -0.27 (0.48) |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 381
  Week 36 | -0.25 (0.48) | -0.43 (0.60) | -0.52 (0.56)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -0.25 (0.48) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -0.26 (0.48) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | -0.27 (0.48) | -0.42 (0.57) | -0.55 (0.55)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -0.28 (0.50) | -0.43 (0.59) | -0.55 (0.56)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -0.29 (0.51) | -0.44 (0.59) | -0.56 (0.58)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -0.29 (0.51) | -0.45 (0.59) | -0.56 (0.57)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -0.29 (0.50) | -0.42 (0.61) | -0.59 (0.58)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -0.30 (0.48) | -0.40 (0.62) | -0.60 (0.60)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -0.30 (0.49) | -0.48 (0.59) | -0.60 (0.58)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -0.31 (0.50) | -0.49 (0.59) | -0.60 (0.57)
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | -0.33 (0.51) | -0.49 (0.60) | -0.58 (0.53)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -0.33 (0.53) | -0.52 (0.60) | -0.58 (0.55)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -0.31 (0.53) | -0.41 (0.62) | -0.51 (0.50)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -0.32 (0.56) | -0.29 (0.69) | -0.52 (0.48)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -0.32 (0.53) | -0.25 (0.68) | -0.44 (0.58)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -0.32 (0.53) | -0.75 (NA) — SD not estimable as there is only one participant. | -0.75 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -0.35 (0.57) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -0.34 (0.58) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -0.31 (0.61) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -0.35 (0.55) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -0.32 (0.57) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -0.36 (0.56) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -0.34 (0.59) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -0.35 (0.59) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -0.37 (0.59) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -0.35 (0.54) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -0.31 (0.60) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -0.29 (0.62) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -0.41 (0.58) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -0.88 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | -0.22 (0.62) | -0.37 (0.63) | -0.51 (0.62)
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | -0.08 (0.63) | -0.17 (0.62) | -0.28 (0.73)

34. Secondary Outcome: Percentage of Participants Achieving HAQ-DI Decrease From Baseline of at Least 0.22 Through Week 372
Description: as for outcome 32
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 35.0 | 59.2 | 67.0
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | 37.0 |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 40.7 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 41.7 |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | 48.0 | 61.5 | 65.7
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 51.0 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 49.5 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 50.3 | 59.9 | 68.3
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 54.3 |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | 50.0 |  |
  Week 36: number analyzed (Participants) | 172 | 206 | 381
  Week 36 | 48.3 | 55.8 | 71.4
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 48.8 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 50.9 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 50.3 | 58.2 | 70.6
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | 54.1 | 59.7 | 71.9
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | 54.0 | 59.6 | 69.9
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | 53.6 | 63.3 | 69.5
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 51.8 | 57.2 | 73.9
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | 54.9 | 56.7 | 73.8
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 52.3 | 62.8 | 73.2
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | 53.2 | 57.8 | 74.9
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 55.8 | 61.9 | 75.0
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | 53.8 | 70.0 | 76.4
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 53.4 | 62.2 | 69.7
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | 57.0 | 47.6 | 71.7
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 55.0 | 50.0 | 59.1
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | 51.4 | 100.0 | 100.0
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 55.8 |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | 52.0 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 50.5 |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | 54.4 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 50.0 |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | 54.7 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 47.6 |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | 54.3 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 51.9 |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | 51.6 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 50.9 |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | 47.5 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 62.5 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 100.0 |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | 46.8 | 55.4 | 68.9
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | 44.6 | 44.6 | 56.2

35. Secondary Outcome: Change From Baseline of Preceding Study in Physician's Global Assessment of Arthritis (PGA) Through Week 372
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm visual analog scale where 0 = very well and 100 = very poorly.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | -10.77 (21.64) | -41.57 (22.92) | -43.09 (23.21)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -13.48 (20.82) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -16.78 (21.81) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -20.59 (23.69) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | -24.33 (23.00) | -40.22 (23.50) | -42.77 (23.09)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -26.64 (22.86) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -27.12 (23.28) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | -27.56 (23.81) | -40.65 (24.02) | -43.81 (23.23)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -29.22 (24.18) |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | -27.80 (24.05) |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | -29.94 (22.82) | -41.60 (24.88) | -44.81 (21.41)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -31.58 (21.55) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -31.60 (22.50) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | -33.04 (23.41) | -41.92 (23.36) | -45.71 (21.52)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -32.82 (24.00) | -41.84 (23.31) | -45.20 (22.00)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -33.68 (24.19) | -42.48 (22.83) | -47.05 (21.35)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -33.39 (25.87) | -41.31 (25.12) | -46.42 (22.33)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -34.12 (23.79) | -43.26 (24.46) | -47.35 (21.98)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -35.70 (24.63) | -43.55 (23.34) | -48.04 (22.43)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -35.14 (25.13) | -45.11 (23.65) | -46.99 (22.76)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -37.24 (25.90) | -45.51 (24.94) | -47.50 (20.77)
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | -39.11 (24.31) | -45.70 (27.19) | -45.85 (22.35)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -37.72 (24.91) | -48.04 (25.43) | -46.65 (21.24)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -39.55 (24.87) | -45.54 (24.77) | -45.07 (22.38)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -37.34 (25.47) | -44.62 (29.00) | -46.01 (20.30)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -39.13 (24.79) | -33.75 (36.86) | -44.50 (19.39)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -40.46 (22.73) | -30.00 (NA) — SD not estimable as there is only one participant. | -53.50 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -40.80 (23.52) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -40.08 (23.25) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -41.67 (24.00) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -41.55 (23.74) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -41.13 (24.71) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -42.46 (22.75) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -42.21 (25.60) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -41.40 (22.39) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -42.18 (22.71) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -42.73 (22.93) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -39.55 (25.31) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -38.71 (24.27) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -40.25 (18.36) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -47.00 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 222 | 412
  EOT | -30.72 (27.55) | -39.86 (26.19) | -45.04 (24.76)
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | -20.31 (26.25) | -30.01 (25.67) | -36.11 (27.05)

36. Secondary Outcome: Change From Baseline of Preceding Study in Subject's Global Assessment of Arthritis (SGA) Through Week 372
Description: The participant assessed his/her own disease activity on a VAS of 0-100 mm on the questionnaire form. Higher SGA (100 mm VAS) scores indicate greater activity impairment.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | -6.82 (25.41) | -37.24 (29.85) | -35.60 (26.98)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -11.31 (24.37) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -13.42 (25.21) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -17.89 (27.08) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | -20.60 (26.15) | -36.80 (30.55) | -34.81 (27.68)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -23.45 (27.01) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -24.35 (27.63) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | -24.78 (26.98) | -37.13 (30.97) | -36.25 (27.07)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -27.29 (27.34) |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | -27.78 (28.04) |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | -27.45 (27.10) | -37.33 (30.74) | -37.57 (25.19)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -29.23 (27.43) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -29.01 (27.10) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | -29.80 (27.43) | -36.12 (29.92) | -37.40 (26.38)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -30.39 (28.54) | -36.18 (30.34) | -37.46 (26.55)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -31.18 (28.44) | -36.86 (29.67) | -38.42 (25.49)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -29.73 (30.45) | -35.33 (31.10) | -38.26 (25.81)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -32.65 (30.12) | -35.75 (30.98) | -38.50 (27.57)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -31.75 (30.27) | -35.54 (31.35) | -39.69 (26.38)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -31.87 (29.95) | -38.88 (29.82) | -39.56 (27.28)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -32.61 (31.77) | -38.66 (30.54) | -37.79 (27.53)
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | -33.67 (29.23) | -38.99 (31.62) | -37.44 (27.31)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -34.15 (30.71) | -39.62 (29.17) | -38.45 (26.52)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -33.59 (30.34) | -38.36 (28.96) | -38.89 (26.37)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -33.56 (30.55) | -38.41 (32.82) | -38.41 (25.29)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -34.94 (29.42) | -49.90 (33.93) | -42.09 (25.39)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -35.65 (29.79) | -83.50 (NA) — SD not estimable as there is only one participant. | -57.00 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -33.69 (32.20) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -34.81 (32.30) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -35.14 (31.35) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -34.84 (31.90) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -34.57 (33.12) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -36.39 (30.81) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -35.51 (32.04) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -36.97 (33.07) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -37.52 (30.54) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -35.50 (30.28) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -33.11 (29.66) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -28.87 (31.14) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -40.29 (28.74) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -71.50 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 223 | 412
  EOT | -26.04 (31.99) | -33.53 (32.73) | -36.57 (28.95)
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | -18.67 (29.38) | -27.86 (33.15) | -22.79 (30.38)

37. Secondary Outcome: Change From Baseline of Preceding Study in Subject's Global Assessment of Arthritis Pain (SGAP) Through Week 372
Description: The participant assessed his/her own pain severity on a visual analog scale (VAS) of 0-100 mm on the questionnaire form. Higher SGA of pain (100 mm VAS) scores indicated greater activity pain.
Time Frame: as for outcome 8
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | -7.37 (25.85) | -36.09 (30.09) | -34.79 (26.98)
  Week 2: number analyzed (Participants) | 200 | 0 | 0
  Week 2 | -11.21 (23.60) |  |
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | -13.10 (24.45) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | -17.70 (26.93) |  |
  Week 12: number analyzed (Participants) | 198 | 218 | 408
  Week 12 | -20.54 (25.98) | -35.75 (30.36) | -34.27 (28.19)
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | -23.12 (26.94) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | -24.00 (27.30) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | -24.41 (26.68) | -36.38 (30.17) | -36.17 (27.15)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | -26.74 (27.81) |  |
  Week 32: number analyzed (Participants) | 179 | 0 | 0
  Week 32 | -27.41 (28.35) |  |
  Week 36: number analyzed (Participants) | 172 | 205 | 381
  Week 36 | -26.73 (28.04) | -36.68 (30.38) | -37.30 (26.59)
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | -28.62 (28.43) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | -29.08 (27.27) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | -30.08 (27.09) | -35.88 (30.24) | -37.16 (26.89)
  Week 60: number analyzed (Participants) | 157 | 191 | 356
  Week 60 | -30.88 (28.64) | -35.77 (30.45) | -36.93 (27.51)
  Week 72: number analyzed (Participants) | 150 | 183 | 349
  Week 72 | -30.47 (28.23) | -36.54 (29.83) | -37.36 (26.86)
  Week 84: number analyzed (Participants) | 140 | 180 | 338
  Week 84 | -29.41 (31.51) | -35.14 (30.67) | -37.58 (27.07)
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | -31.59 (31.98) | -34.55 (30.47) | -37.83 (27.59)
  Week 108: number analyzed (Participants) | 133 | 164 | 267
  Week 108 | -31.16 (31.19) | -35.52 (30.77) | -38.72 (26.97)
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | -31.92 (30.85) | -38.32 (29.85) | -38.34 (27.88)
  Week 132: number analyzed (Participants) | 126 | 116 | 175
  Week 132 | -32.42 (31.62) | -38.30 (29.75) | -36.66 (26.60)
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | -33.53 (31.99) | -39.02 (29.85) | -36.34 (25.75)
  Week 156: number analyzed (Participants) | 119 | 70 | 106
  Week 156 | -33.61 (31.76) | -40.11 (29.13) | -37.08 (26.55)
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | -34.24 (32.17) | -38.27 (28.57) | -36.96 (26.23)
  Week 180: number analyzed (Participants) | 114 | 21 | 46
  Week 180 | -33.40 (32.56) | -42.90 (30.70) | -37.85 (25.95)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | -34.50 (30.26) | -50.81 (36.83) | -40.86 (28.24)
  Week 204: number analyzed (Participants) | 107 | 1 | 1
  Week 204 | -35.88 (30.63) | -82.50 (NA) — SD not estimable as there is only one participant. | -58.00 (NA) — SD not estimable as there is only one participant.
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | -33.21 (33.60) |  |
  Week 228: number analyzed (Participants) | 98 | 0 | 0
  Week 228 | -34.44 (33.92) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | -34.98 (32.39) |  |
  Week 252: number analyzed (Participants) | 90 | 0 | 0
  Week 252 | -34.88 (33.20) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | -34.81 (34.02) |  |
  Week 276: number analyzed (Participants) | 86 | 0 | 0
  Week 276 | -36.12 (32.40) |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | -34.63 (33.46) |  |
  Week 300: number analyzed (Participants) | 81 | 0 | 0
  Week 300 | -35.73 (34.47) |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | -35.42 (33.21) |  |
  Week 324: number analyzed (Participants) | 64 | 0 | 0
  Week 324 | -33.43 (34.58) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | -32.56 (32.27) |  |
  Week 348: number analyzed (Participants) | 40 | 0 | 0
  Week 348 | -25.96 (33.18) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | -35.59 (26.94) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -58.60 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 223 | 412
  EOT | -26.57 (32.59) | -33.82 (32.32) | -35.84 (30.02)
  EOS: number analyzed (Participants) | 101 | 65 | 89
  EOS | -19.77 (28.17) | -29.87 (31.05) | -21.54 (30.66)

38. Secondary Outcome: Change From Baseline of Preceding Study in Short Form Health Survey - 36 Questions, Version 2 (SF-36v2) Physical Component Summary Score Through Week 372
Description: The SF-36v2 was scored for the 8 subscales (each range: 0-100 scale): 1. physical functioning, 2. role physical, 3. bodily pain, 4. general health, 5. vitality, 6. social functioning, 7. role-emotional, and 8. mental health. Physical Component Summary Score, Mental Component Summary Score and Role/Social Component Summary Score were calculated based on the 2007 General Japanese Population Means and Standard Deviations and coefficient. Component summary measures had means of 50 in 2007 General Japanese Population and deviation was expressed by the scale of 10. Higher score indicated better health state.
Time Frame: Baseline of preceding study and weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 216, 228, 240, 252, 264, 276, 288, 300, 312, 324, 336, 348, 360, 372, EOT
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 223 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | -0.55 (13.12) | 11.62 (12.80) | 11.60 (12.48)
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 0.30 (13.81) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 1.53 (12.85) |  |
  Week 12: number analyzed (Participants) | 198 | 0 | 0
  Week 12 | 2.52 (13.47) |  |
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 4.10 (13.36) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 3.72 (14.22) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 3.56 (13.69) | 12.55 (13.84) | 13.23 (12.43)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 3.97 (14.13) |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | 4.14 (13.35) |  |
  Week 36: number analyzed (Participants) | 172 | 0 | 0
  Week 36 | 3.63 (14.08) |  |
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 4.27 (13.92) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 4.49 (13.26) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 4.51 (13.42) | 12.31 (13.60) | 13.52 (12.11)
  Week 60: number analyzed (Participants) | 138 | 0 | 0
  Week 60 | 5.89 (13.46) |  |
  Week 72: number analyzed (Participants) | 149 | 183 | 349
  Week 72 | 4.94 (14.02) | 12.35 (14.10) | 13.48 (13.23)
  Week 84: number analyzed (Participants) | 77 | 0 | 0
  Week 84 | 5.59 (13.30) |  |
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 5.02 (14.20) | 12.15 (14.95) | 14.20 (13.16)
  Week 108: number analyzed (Participants) | 2 | 0 | 0
  Week 108 | 0.27 (14.50) |  |
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 5.01 (14.34) | 12.59 (15.29) | 14.59 (13.37)
  Week 132: number analyzed (Participants) | 1 | 0 | 0
  Week 132 | -7.23 (NA) — SD not estimable as there is only one participant. |  |
  Week 144: number analyzed (Participants) | 120 | 97 | 412
  Week 144 | 6.94 (14.43) | 12.46 (14.20) | 14.38 (13.42)
  Week 156: number analyzed (Participants) | 1 | 0 | 0
  Week 156 | -31.60 (NA) — SD not estimable as there is only one participant. |  |
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 6.46 (15.80) | 9.64 (12.16) | 13.94 (13.97)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 6.43 (14.75) | 10.42 (16.12) | 12.60 (12.95)
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 6.73 (15.24) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 6.13 (16.19) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 5.97 (17.28) |  |
  Week 276: number analyzed (Participants) | 1 | 0 | 0
  Week 276 | -22.64 (NA) — SD not estimable as there is only one participant. |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 6.21 (16.43) |  |
  Week 300: number analyzed (Participants) | 1 | 0 | 0
  Week 300 | 4.73 (NA) — SD not estimable as there is only one participant. |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 6.13 (16.23) |  |
  Week 324: number analyzed (Participants) | 6 | 0 | 0
  Week 324 | 21.10 (23.80) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 4.33 (15.78) |  |
  Week 348: number analyzed (Participants) | 9 | 0 | 0
  Week 348 | -5.21 (13.68) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 6.92 (9.75) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0.16 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 218 | 405
  EOT | 3.44 (NA) — SD not estimable as there is only one participant. | 10.29 (15.46) | 12.62 (13.23)

39. Secondary Outcome: Change From Baseline of Preceding Study in SF-36v2 Mental Component Summary Score Through Week 372
Description: as for outcome 38
Time Frame: as for outcome 38
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 223 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 3.00 (8.40) | 2.94 (8.52) | 2.69 (8.67)
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 3.88 (8.86) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 3.85 (9.51) |  |
  Week 12: number analyzed (Participants) | 198 | 0 | 0
  Week 12 | 4.72 (9.08) |  |
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 4.61 (9.25) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 4.97 (9.18) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 6.01 (9.13) | 2.02 (9.15) | 2.61 (9.04)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 5.38 (9.74) |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | 5.13 (9.20) |  |
  Week 36: number analyzed (Participants) | 172 | 0 | 0
  Week 36 | 5.18 (9.05) |  |
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 5.70 (9.27) |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 5.79 (9.33) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 5.52 (9.24) | 1.74 (8.78) | 2.89 (8.76)
  Week 60: number analyzed (Participants) | 138 | 0 | 0
  Week 60 | 5.27 (9.15) |  |
  Week 72: number analyzed (Participants) | 149 | 183 | 349
  Week 72 | 5.28 (8.83) | 2.87 (9.31) | 2.80 (8.94)
  Week 84: number analyzed (Participants) | 77 | 0 | 0
  Week 84 | 5.58 (9.06) |  |
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 5.42 (9.17) | 2.10 (8.98) | 2.22 (9.52)
  Week 108: number analyzed (Participants) | 2 | 0 | 0
  Week 108 | 3.89 (7.29) |  |
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 4.64 (8.73) | 2.40 (8.67) | 1.62 (9.24)
  Week 132: number analyzed (Participants) | 1 | 0 | 0
  Week 132 | -2.52 (NA) — SD not estimable as there is only one participant. |  |
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 4.38 (9.16) | 1.56 (9.22) | 1.65 (8.15)
  Week 156: number analyzed (Participants) | 1 | 0 | 0
  Week 156 | 2.17 (NA) — SD not estimable as there is only one participant. |  |
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 4.09 (9.41) | 2.41 (8.92) | 2.04 (8.41)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 3.56 (8.52) | 2.23 (3.58) | 2.31 (6.81)
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 2.95 (9.70) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 3.45 (9.60) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 4.03 (9.69) |  |
  Week 276: number analyzed (Participants) | 1 | 0 | 0
  Week 276 | 6.20 (NA) — SD not estimable as there is only one participant. |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 3.72 (9.09) |  |
  Week 300: number analyzed (Participants) | 1 | 0 | 0
  Week 300 | 11.12 (NA) — SD not estimable as there is only one participant. |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 4.62 (10.58) |  |
  Week 324: number analyzed (Participants) | 6 | 0 | 0
  Week 324 | 7.83 (10.42) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 3.78 (8.57) |  |
  Week 348: number analyzed (Participants) | 9 | 0 | 0
  Week 348 | 2.80 (6.90) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 5.15 (9.50) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -3.24 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 218 | 405
  EOT | 3.63 (9.97) | 1.54 (9.91) | 2.16 (9.29)

40. Secondary Outcome: Change From Baseline of Preceding Study in SF-36v2 Role/Social Component Summary Score Through Week 372
Description: as for outcome 38
Time Frame: as for outcome 38
Population: FAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 223 | 412
units on a scale
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | -0.52 (12.29) | 5.21 (13.96) | 5.45 (15.40)
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 0.29 (11.16) |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 1.30 (12.39) |  |
  Week 12: number analyzed (Participants) | 198 | 0 | 0
  Week 12 | 1.70 (12.00) |  |
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 2.84 (11.58) |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 2.33 (12.73) |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 1.59 (11.27) | 5.06 (13.55) | 5.56 (15.36)
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 2.68 (11.73) |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | 3.75 (11.55) |  |
  Week 36: number analyzed (Participants) | 172 | 0 | 0
  Week 36 | 1.66 (12.08) |  |
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 2.42 (12.57) |  |
  Week 44: number analyzed (Participants) | 172 | 0 | 0
  Week 44 | 1.93 (12.08) |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 2.85 (11.64) | 5.06 (14.54) | 5.80 (15.27)
  Week 60: number analyzed (Participants) | 138 | 0 | 0
  Week 60 | 3.05 (12.65) |  |
  Week 72: number analyzed (Participants) | 149 | 183 | 349
  Week 72 | 2.56 (12.84) | 5.65 (13.93) | 6.37 (15.33)
  Week 84: number analyzed (Participants) | 77 | 0 | 0
  Week 84 | 0.81 (12.75) |  |
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 2.67 (12.51) | 4.30 (13.56) | 5.80 (15.61)
  Week 108: number analyzed (Participants) | 2 | 0 | 0
  Week 108 | -1.62 (1.64) |  |
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 2.97 (12.90) | 4.55 (14.28) | 5.92 (16.32)
  Week 132: number analyzed (Participants) | 1 | 0 | 0
  Week 132 | -5.25 (NA) — SD not estimable as there is only one participant. |  |
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 2.64 (12.95) | 5.18 (14.52) | 5.43 (15.59)
  Week 156: number analyzed (Participants) | 1 | 0 | 0
  Week 156 | 5.75 (NA) — SD not estimable as there is only one participant. |  |
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 2.88 (12.83) | 0.50 (12.86) | 4.11 (14.33)
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 2.75 (12.81) | -0.97 (12.36) | 2.17 (15.20)
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 3.50 (13.80) |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 3.46 (13.20) |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 2.65 (13.28) |  |
  Week 276: number analyzed (Participants) | 1 | 0 | 0
  Week 276 | 1.82 (NA) — SD not estimable as there is only one participant. |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 3.99 (12.95) |  |
  Week 300: number analyzed (Participants) | 1 | 0 | 0
  Week 300 | 12.34 (NA) — SD not estimable as there is only one participant. |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 3.87 (14.89) |  |
  Week 324: number analyzed (Participants) | 6 | 0 | 0
  Week 324 | 15.79 (12.43) |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 3.54 (13.56) |  |
  Week 348: number analyzed (Participants) | 9 | 0 | 0
  Week 348 | -1.11 (12.48) |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 1.64 (12.72) |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | -8.61 (NA) — SD not estimable as there is only one participant. |  |
  EOT: number analyzed (Participants) | 201 | 218 | 405
  EOT | 2.06 (14.35) | 3.92 (13.85) | 4.74 (16.31)

41. Secondary Outcome: Percentage of Participants Achieving SF-36v2 Physical Component Summary Score of Difference >= 5 Through Week 372
Description: as for outcome 38
Time Frame: Baseline of preceding study and weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 216, 240, 252, 264, 276, 288, 300, 312, 324, 336, 348, 360, 372, EOT
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 223 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 34.0 | 70 | 71.1
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 33.7 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 40.2 |  |
  Week 12: number analyzed (Participants) | 198 | 0 | 0
  Week 12 | 39.4 |  |
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 43.4 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 40.0 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 44.4 | 70.5 | 74.1
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 42.9 |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | 44.4 |  |
  Week 36: number analyzed (Participants) | 172 | 0 | 0
  Week 36 | 45.3 |  |
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 47.0 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 47.2 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 45.4 | 73.0 | 74.7
  Week 60: number analyzed (Participants) | 138 | 0 | 0
  Week 60 | 47.8 |  |
  Week 72: number analyzed (Participants) | 149 | 183 | 349
  Week 72 | 47.7 | 68.3 | 73.9
  Week 84: number analyzed (Participants) | 77 | 0 | 0
  Week 84 | 50.6 |  |
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 43.8 | 71.7 | 75.9
  Week 108: number analyzed (Participants) | 2 | 0 | 0
  Week 108 | 50.0 |  |
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 44.6 | 68.2 | 79.3
  Week 132: number analyzed (Participants) | 1 | 0 | 0
  Week 132 | 0 |  |
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 53.3 | 66.0 | 82.4
  Week 156: number analyzed (Participants) | 1 | 0 | 0
  Week 156 | 0 |  |
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 50.0 | 70.3 | 77.6
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 52.3 | 62.5 | 77.3
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 51.9 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 53.7 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 52.2 |  |
  Week 276: number analyzed (Participants) | 1 | 0 | 0
  Week 276 | 0 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 48.8 |  |
  Week 300: number analyzed (Participants) | 1 | 0 | 0
  Week 300 | 0 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 48.1 |  |
  Week 324: number analyzed (Participants) | 6 | 0 | 0
  Week 324 | 66.7 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 43.4 |  |
  Week 348: number analyzed (Participants) | 9 | 0 | 0
  Week 348 | 11.1 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 56.3 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0 |  |
  EOT: number analyzed (Participants) | 201 | 218 | 405
  EOT | 41.8 | 61.0 | 306

42. Secondary Outcome: Percentage of Participants Achieving SF-36v2 Mental Component Summary Score of Difference >= 5 Through Week 372
Description: as for outcome 38
Time Frame: as for outcome 41
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 223 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 43.0 | 39.9 | 37.4
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 42.7 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 47.2 |  |
  Week 12: number analyzed (Participants) | 198 | 0 | 0
  Week 12 | 43.4 |  |
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 45.4 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 45.3 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 51.9 | 37.2 | 37.6
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 47.8 |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | 48.3 |  |
  Week 36: number analyzed (Participants) | 172 | 0 | 0
  Week 36 | 47.7 |  |
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 49.4 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 49.1 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 51.5 | 33.2 | 39.2
  Week 60: number analyzed (Participants) | 138 | 0 | 0
  Week 60 | 48.6 |  |
  Week 72: number analyzed (Participants) | 149 | 183 | 349
  Week 72 | 53.7 | 39.3 | 35.8
  Week 84: number analyzed (Participants) | 77 | 0 | 0
  Week 84 | 57.1 |  |
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 49.6 | 33.5 | 38.4
  Week 108: number analyzed (Participants) | 2 | 0 | 0
  Week 108 | 50.0 |  |
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 45.4 | 37.2 | 33.8
  Week 132: number analyzed (Participants) | 1 | 0 | 0
  Week 132 | 0 |  |
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 47.5 | 30.9 | 28.7
  Week 156: number analyzed (Participants) | 1 | 0 | 0
  Week 156 | 0 |  |
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 41.4 | 32.4 | 34.2
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 39.6 | 37.5 | 31.8
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 37.5 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 42.1 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 43.3 |  |
  Week 276: number analyzed (Participants) | 1 | 0 | 0
  Week 276 | 100 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 41.7 |  |
  Week 300: number analyzed (Participants) | 1 | 0 | 0
  Week 300 | 100 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 43.0 |  |
  Week 324: number analyzed (Participants) | 6 | 0 | 0
  Week 324 | 33.3 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 37.7 |  |
  Week 348: number analyzed (Participants) | 9 | 0 | 0
  Week 348 | 22.2 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 43.8 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0 |  |
  EOT: number analyzed (Participants) | 201 | 218 | 405
  EOT | 39.8 | 35.8 | 34.6

43. Secondary Outcome: Percentage of Participants Achieving SF-36v2 Role/Social Component Summary Score of Difference >= 5 Through Week 372
Description: as for outcome 38
Time Frame: as for outcome 41
Population: FAS population with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 223 | 412
percentage of participants
  Week 0: number analyzed (Participants) | 200 | 223 | 412
  Week 0 | 26.0 | 44.8 | 48.5
  Week 4: number analyzed (Participants) | 199 | 0 | 0
  Week 4 | 27.6 |  |
  Week 8: number analyzed (Participants) | 199 | 0 | 0
  Week 8 | 35.7 |  |
  Week 12: number analyzed (Participants) | 198 | 0 | 0
  Week 12 | 39.9 |  |
  Week 16: number analyzed (Participants) | 196 | 0 | 0
  Week 16 | 39.8 |  |
  Week 20: number analyzed (Participants) | 190 | 0 | 0
  Week 20 | 38.4 |  |
  Week 24: number analyzed (Participants) | 187 | 207 | 394
  Week 24 | 36.4 | 47.8 | 48.0
  Week 28: number analyzed (Participants) | 184 | 0 | 0
  Week 28 | 39.1 |  |
  Week 32: number analyzed (Participants) | 180 | 0 | 0
  Week 32 | 40.0 |  |
  Week 36: number analyzed (Participants) | 172 | 0 | 0
  Week 36 | 33.1 |  |
  Week 40: number analyzed (Participants) | 168 | 0 | 0
  Week 40 | 38.7 |  |
  Week 44: number analyzed (Participants) | 163 | 0 | 0
  Week 44 | 38.7 |  |
  Week 48: number analyzed (Participants) | 163 | 196 | 367
  Week 48 | 40.5 | 46.4 | 47.1
  Week 60: number analyzed (Participants) | 138 | 0 | 0
  Week 60 | 39.9 |  |
  Week 72: number analyzed (Participants) | 149 | 183 | 349
  Week 72 | 38.9 | 47.5 | 46.7
  Week 84: number analyzed (Participants) | 77 | 0 | 0
  Week 84 | 29.9 |  |
  Week 96: number analyzed (Participants) | 137 | 173 | 307
  Week 96 | 38.7 | 42.8 | 48.2
  Week 108: number analyzed (Participants) | 2 | 0 | 0
  Week 108 | 0 |  |
  Week 120: number analyzed (Participants) | 130 | 148 | 213
  Week 120 | 39.2 | 45.3 | 49.3
  Week 132: number analyzed (Participants) | 1 | 0 | 0
  Week 132 | 0 |  |
  Week 144: number analyzed (Participants) | 120 | 97 | 136
  Week 144 | 38.3 | 51.5 | 48.5
  Week 156: number analyzed (Participants) | 1 | 0 | 0
  Week 156 | 100 |  |
  Week 168: number analyzed (Participants) | 116 | 37 | 76
  Week 168 | 39.7 | 35.1 | 40.8
  Week 192: number analyzed (Participants) | 111 | 8 | 22
  Week 192 | 38.7 | 25.0 | 31.8
  Week 216: number analyzed (Participants) | 104 | 0 | 0
  Week 216 | 40.0 |  |
  Week 240: number analyzed (Participants) | 95 | 0 | 0
  Week 240 | 41.1 |  |
  Week 264: number analyzed (Participants) | 90 | 0 | 0
  Week 264 | 37.8 |  |
  Week 276: number analyzed (Participants) | 1 | 0 | 0
  Week 276 | 0 |  |
  Week 288: number analyzed (Participants) | 84 | 0 | 0
  Week 288 | 42.9 |  |
  Week 300: number analyzed (Participants) | 1 | 0 | 0
  Week 300 | 100.0 |  |
  Week 312: number analyzed (Participants) | 79 | 0 | 0
  Week 312 | 45.6 |  |
  Week 324: number analyzed (Participants) | 6 | 0 | 0
  Week 324 | 83.3 |  |
  Week 336: number analyzed (Participants) | 53 | 0 | 0
  Week 336 | 39.6 |  |
  Week 348: number analyzed (Participants) | 9 | 0 | 0
  Week 348 | 22.2 |  |
  Week 360: number analyzed (Participants) | 16 | 0 | 0
  Week 360 | 31.3 |  |
  Week 372: number analyzed (Participants) | 1 | 0 | 0
  Week 372 | 0.0 |  |
  EOT: number analyzed (Participants) | 201 | 218 | 405
  EOT | 39.8 | 43.1 | 44.7

44. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy
Description: Participants who discontinued due to lack of efficacy have been reported.
Time Frame: Baseline up to week 372
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
Number analyzed (Participants) | 201 | 224 | 412
percentage of participants | 19.4 | 4.9 | 3.4

ADVERSE EVENTS:
Time Frame: Baseline up to EOS (Up to 376 weeks)
Description: Safety Population
Arm/Group | Participants Who Completed 015K-CL-RAJ1 | Participants Who Completed 015K-CL-RAJ3 | Participants Who Completed 015K-CL-RAJ4
All-Cause Mortality (participants affected / at risk) | 0/201 | 1/225 | 1/417
Serious Adverse Events (participants affected / at risk) | 59/201 | 56/225 | 84/417
Other Adverse Events (participants affected / at risk) | 181/201 | 174/225 | 358/417
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Completed 015K-CL-RAJ1 (N=201) | Participants Who Completed 015K-CL-RAJ3 (N=225) | Participants Who Completed 015K-CL-RAJ4 (N=417)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Urachal abnormality (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Steroid withdrawal syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Maculopathy (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 3 (3)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dacryocystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 4 (4) | 9 (9)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Keratitis herpetic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 6 (6) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fractured ischium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 4 (5) | 1 (1) | 4 (4)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2)
Bronchoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Endoscopy large bowel (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 0 (0)
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Extraskeletal chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 2 (2)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ankle operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Jaw operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve neurostimulation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Completed 015K-CL-RAJ1 (N=201) | Participants Who Completed 015K-CL-RAJ3 (N=225) | Participants Who Completed 015K-CL-RAJ4 (N=417)
Dry eye (Eye disorders) | 12 (13) | 3 (3) | 5 (5)
Constipation (Gastrointestinal disorders) | 21 (23) | 14 (15) | 25 (27)
Dental caries (Gastrointestinal disorders) | 19 (24) | 13 (16) | 29 (38)
Diarrhoea (Gastrointestinal disorders) | 16 (18) | 9 (16) | 12 (14)
Gastritis (Gastrointestinal disorders) | 12 (12) | 8 (8) | 7 (7)
Nausea (Gastrointestinal disorders) | 12 (13) | 11 (11) | 18 (22)
Periodontitis (Gastrointestinal disorders) | 13 (16) | 9 (9) | 13 (14)
Hepatic function abnormal (Hepatobiliary disorders) | 7 (8) | 7 (8) | 27 (27)
Bronchitis (Infections and infestations) | 29 (76) | 22 (30) | 28 (32)
Cystitis (Infections and infestations) | 17 (35) | 17 (25) | 27 (50)
Gastroenteritis (Infections and infestations) | 24 (30) | 16 (17) | 22 (30)
Herpes zoster (Infections and infestations) | 35 (36) | 35 (36) | 63 (68)
Influenza (Infections and infestations) | 35 (41) | 22 (23) | 44 (51)
Nasopharyngitis (Infections and infestations) | 110 (368) | 91 (211) | 195 (423)
Pharyngitis (Infections and infestations) | 22 (65) | 14 (33) | 33 (57)
Upper respiratory tract infection (Infections and infestations) | 23 (76) | 15 (26) | 26 (38)
Contusion (Injury, poisoning and procedural complications) | 22 (26) | 17 (19) | 35 (39)
Blood creatine phosphokinase increased (Investigations) | 29 (47) | 23 (35) | 45 (55)
Lymphocyte count decreased (Investigations) | 8 (8) | 7 (9) | 28 (49)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (26) | 12 (15) | 28 (30)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 50 (78) | 27 (35) | 55 (61)
Headache (Nervous system disorders) | 16 (27) | 9 (12) | 19 (95)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (28) | 12 (13) | 20 (23)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (24) | 3 (3) | 8 (8)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 9 (13) | 12 (19)
Eczema (Skin and subcutaneous tissue disorders) | 19 (26) | 10 (12) | 13 (17)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 13 (16) | 4 (5) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 12 (17) | 4 (4) | 13 (14)
Hypertension (Vascular disorders) | 30 (30) | 14 (14) | 28 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT01638013/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT01638013/SAP_001.pdf